CLINICAL TRIAL: NCT06433908
Title: A Phase 1, Randomized, Open-label, Single Dose, 2-treatment Arm (200 μg and 800 μg), 4-way Crossover Study in Healthy Participants Aged 18 to 55 to Compare the Pharmacokinetics of Salbutamol Administered Via Metered Dose Inhalers Containing Propellants HFA-152A (Test) and HFA-134A (Reference)
Brief Title: A Study to Compare the Pharmacokinetics (PK) of Salbutamol Administered Via Metered Dose Inhalers (MDI) Containing Propellants HFA-152A (Test) or HFA-134A (Reference) in Healthy Participants Aged 18 to 55 Inclusive
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 219728; 2023-508279-36-00 (Other: EU CT number)
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Asthma; Healthy Participants
Keywords: salbutamol; propellant HFA-152a; propellant HFA-134a; metered dose inhalers; healthy participants; asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: 4-way crossover study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Salbutamol 200 μg (Experimental): Participants will receive single 200 μg doses given as 2x100 μg (ex-valve) at 20-second intervals. The intervention period will be 10 days with dosing with either HFA-152a or HFA-134a on Day 1, Day 4, Day 7, and Day 10.
  Interventions: Drug: Salbutamol HFA-152a; Drug: Salbutamol HFA-134a
- Cohort 2: Salbutamol 800 μg (Experimental): Participants will receive single 800 μg doses given as 8x100 μg (ex-valve) at 20-second intervals. The intervention period will be 10 days with dosing with either HFA-152a or HFA-134a on Day 1, Day 4, Day 7, and Day 10.
  Interventions: Drug: Salbutamol HFA-152a; Drug: Salbutamol HFA-134a

INTERVENTIONS:
Drug: Salbutamol HFA-152a — 100 µg (ex-valve), given at 20-second intervals.
Drug: Salbutamol HFA-134a — 100 µg (ex-valve), given at 20-second intervals.

SUMMARY:
The primary objective of the study is to characterize the PK of single doses of salbutamol in healthy participants delivered via an MDI containing propellant HFA-152a (test), and to compare with an MDI containing propellant HFA-134a (reference).

ELIGIBILITY:
Inclusion Criteria:

1. Sex: male or female; females may be of childbearing potential, of nonchild bearing potential, or postmenopausal.
2. Age: 18 to 55 years inclusive.
3. Weight: 45 to 110 kg inclusive
4. Status: healthy participants.
5. Females must not be pregnant or lactating.
6. All prescribed medication must have been stopped at least 30 days prior to admission to the clinical research center based on investigator judgment. An exception is made for hormonal contraceptives, which may be used throughout the study.
7. All over-the-counter medication, vitamin preparations and other food supplements, or herbal medications (e.g., St. John's wort) must have been stopped at least 14 days prior to admission to the clinical research center based on investigator judgment. An exception is made for acetaminophen, which is allowed up to admission to the clinical research center.
8. Ability and willingness to abstain from alcohol from 48 hours (2 days) prior to screening, and from 48 hours (2 days) prior to admission until discharge from the clinical research center.
9. Ability and willingness to abstain from methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, energy drinks) from 48 hours (2 days) prior to admission until discharge from the clinical research center.
10. Good physical and mental health on the basis of medical history, physical examination, clinical laboratory, ECG, and vital signs, as judged by the investigator.
11. Serum potassium and serum glucose levels within reference ranges of the clinical research center.
12. Willing and able to sign the informed consent form.
13. Spirometry at screening demonstrating forced expiratory volume ≥80% predicted.

Exclusion Criteria:

1. History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs.
2. History or presence of any form of asthma, including childhood asthma and exercise induced asthma.
3. At screening, systolic blood pressure <90 mmHg or >140 mmHg, or diastolic blood pressure <50 mmHg or >90 mmHg.
4. History of pathological tachycardia, or a pulse rate > 85 beats per minute (bpm) at screening or Day-1.
5. Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
6. Breast cancer within the past 10 years.
7. A QTcF value of >450 msec at screening based on a triplicate measurement taken at a single timepoint.
8. Vaccine(s) within 2 weeks prior to admission, or plans to receive such vaccines during the study.
9. Donation or loss of more than 450 mL of blood within 60 days prior to (the first) drug administration. Donation or loss of more than 1.5 L of blood (for male participants) or more than 1.0 L of blood (for female participants) in the 10 months prior to (the first) drug administration in the current study.
10. Participation in a drug study within 30 days prior to (the first) drug administration in the current study. Participation in 4 or more other drug studies in the 12 months prior to (the first) drug administration in the current study.
11. Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
12. Presence of hepatitis B surface antigen at screening or within 3 months prior to first dose of study intervention.
13. Positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention. NOTE: Participants with positive hepatitis C antibody test result due to prior resolved disease can be enrolled if a confirmatory negative hepatitis C RNA test is obtained.
14. Positive pre-study drug/alcohol screen, including tetrahydrocannabinol.
15. Positive HIV antibody test.
16. Cotinine levels indicative of smoking or history or use of tobacco- or nicotine containing products within 6 months prior to screening.

    Assessment as ineligible by the investigator based on the results of the clinical laboratory tests or other assessments.
17. Average intake of more than 24 units of alcohol per week: 1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine, or 35 mL of spirits.
18. Regular use of known drugs of abuse, including tetrahydrocannabinol.
19. Use of combustible tobacco products, and non-combustible nicotine delivery systems, inclusive of cigarettes, cigars, pipes, and materials used to "vape" within 6 months prior to screening.
20. Use of any products intended to treat medical conditions that are not approved by the governing health authority in a given country or region (for example, herbal medicine, health supplements, traditional medicine, homeopathic remedies, etc.).
21. Impairment which would prevent the correct and consistent use of an MDI, as determined by the investigator/delegate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of two cohorts: Cohort 1 (200 µg dose) and Cohort 2 (800 µg dose). Each cohort included two treatment sequences, "TRRT" and "RTTR," where T represents salbutamol delivered using HFA-152a MDI (test) and R represents salbutamol delivered using HFA-134a MDI (reference). Participants were randomized to 1 of the 2 treatment sequences within each cohort.
Groups:
- Cohort 1: TRRT1: Healthy participants in Cohort 1 received TRRT1, where "T" represents Salbutamol Hydrofluoroalkane (HFA)-152a (Test) via metered dose inhalers (MDI) as a single 200 ug (2 x 100 µg) administered at 20-second intervals on Day 1, Day 10 and "R" represents Salbutamol HFA-134a (Reference) via MDI as a single 200 ug (2 x 100 µg), administered at 20-second intervals on Day 4, Day 7
- Cohort 1: RTTR1: Healthy participants in Cohort 1 received RTTR1, where "T" represents Salbutamol Hydrofluoroalkane (HFA)-152a (Test) via metered dose inhalers (MDI) as a single 200 ug (2 x 100 µg) administered at 20-second intervals on Day 4, Day 7 and "R" represents Salbutamol HFA-134a (Reference) via MDI as a single 200 ug (2 x 100 µg), administered at 20-second intervals on Day 1, Day 10
- Cohort 2: TRRT2: Healthy participants in Cohort 2 received TRRT2, where "T" represents Salbutamol Hydrofluoroalkane (HFA)-152a (Test) via metered dose inhalers (MDI) as a single 800 ug (8 x 100 µg) administered at 20-second intervals on Day 1, Day 10 and "R" represents Salbutamol HFA-134a (Reference) via MDI as a single 800 ug (8 x 100 µg), administered at 20-second intervals on Day 4, Day 7
- Cohort 2: RTTR2: Healthy participants in Cohort 2 received RTTR2, where "T" represents Salbutamol Hydrofluoroalkane (HFA)-152a (Test) via metered dose inhalers (MDI) as a single 800 ug (8 x 100 µg) administered at 20-second intervals on Day 4, Day 7 and "R" represents Salbutamol HFA-134a (Reference) via MDI as a single 800 ug (8 x 100 µg), administered at 20-second intervals on Day 1, Day 10
Period: Cohort 1 - Treatment Period 1 (Day 1)
Arm/Group | Cohort 1: TRRT1 | Cohort 1: RTTR1 | Cohort 2: TRRT2 | Cohort 2: RTTR2
Started | 16 | 14 | 0 | 0
Completed | 16 | 14 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 1 - Treatment Period 2 (Day 4)
Arm/Group | Cohort 1: TRRT1 | Cohort 1: RTTR1 | Cohort 2: TRRT2 | Cohort 2: RTTR2
Started | 16 | 14 | 0 | 0
Completed | 16 | 14 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 1 - Treatment Period 3 (Day 7)
Arm/Group | Cohort 1: TRRT1 | Cohort 1: RTTR1 | Cohort 2: TRRT2 | Cohort 2: RTTR2
Started | 16 | 14 | 0 | 0
Completed | 15 | 13 | 0 | 0
Not Completed | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Period: Cohort 1 - Treatment Period 4 (Day 10)
Arm/Group | Cohort 1: TRRT1 | Cohort 1: RTTR1 | Cohort 2: TRRT2 | Cohort 2: RTTR2
Started | 15 | 13 | 0 | 0
Completed | 15 | 13 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 2 - Treatment Period 1 (Day 1)
Arm/Group | Cohort 1: TRRT1 | Cohort 1: RTTR1 | Cohort 2: TRRT2 | Cohort 2: RTTR2
Started | 0 | 0 | 14 | 16
Completed | 0 | 0 | 14 | 16
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 2 - Treatment Period 2 (Day 4)
Arm/Group | Cohort 1: TRRT1 | Cohort 1: RTTR1 | Cohort 2: TRRT2 | Cohort 2: RTTR2
Started | 0 | 0 | 14 | 16
Completed | 0 | 0 | 13 | 16
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Period: Cohort 2 - Treatment Period 3 (Day 7)
Arm/Group | Cohort 1: TRRT1 | Cohort 1: RTTR1 | Cohort 2: TRRT2 | Cohort 2: RTTR2
Started | 0 | 0 | 13 | 16
Completed | 0 | 0 | 13 | 16
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 2 - Treatment Period 4 (Day 10)
Arm/Group | Cohort 1: TRRT1 | Cohort 1: RTTR1 | Cohort 2: TRRT2 | Cohort 2: RTTR2
Started | 0 | 0 | 13 | 16
Completed | 0 | 0 | 13 | 16
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: TRRT1 | Cohort 1: RTTR1 | Cohort 2: TRRT2 | Cohort 2: RTTR2 | Total
Number analyzed (Participants) | 16 | 14 | 14 | 16 | 60
Age, Customized [Count of Participants; unit: Participants]
  18 to 55 years | 16 | 14 | 14 | 16 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 10 | 5 | 33
  Male | 5 | 7 | 4 | 11 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 13 | 14 | 13 | 16 | 56
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Cohort 1: Time to Reach Cmax (Tmax)
Description: Blood samples were collected for the analysis of PK parameters.
Time Frame: At pre-dose, 3, 5, 10, 15, 20, 30, and 45 minutes post-dose and at 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose on Day 1 (Period 1), Day 4 (Period 2), Day 7 (Period 3) and Day 10 (Period 4)
Population: Pharmacokinetic Population. "Overall Number of Participants Analyzed" included the total number of participants in Cohort 1. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Median (Full Range); unit: Hour (h)
Groups:
- Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test): Healthy participants in cohort 1 received Salbutamol HFA-152a (Test) via MDI as single dose of 200 ug as inhalation suspension at 20 second intervals administered on Day 1 and Day 10 in the first sequence (TRRT) and Day 4 and Day 7 in the second sequence (RTTR), where T is salbutamol HFA-152a (test) and R is salbutamol HFA-134a (reference).
- Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference): Healthy participants in cohort 1 received Salbutamol HFA-134a (Reference) via MDI as single dose of 200 ug as inhalation suspension at 20 second intervals administered on Day 4 and Day 7 in the first sequence (TRRT) and Day 1 and Day 10 in the second sequence (RTTR), where R is salbutamol HFA-134a (reference) and T is salbutamol HFA-152a (test).
Arm/Group | Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) | Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference)
Number analyzed (Participants) | 30 | 30
Hour (h)
  Day 1: number analyzed (Participants) | 16 | 14
  Day 1 | 2.00 [0.3 to 3.0] | 2.0 [0.8 to 5.0]
  Day 4: number analyzed (Participants) | 14 | 16
  Day 4 | 1.25 [0.3 to 5.0] | 1.00 [0.1 to 3.0]
  Day 7: number analyzed (Participants) | 13 | 15
  Day 7 | 1.50 [0.2 to 4.0] | 1.50 [0.1 to 4.0]
  Day 10: number analyzed (Participants) | 14 | 13
  Day 10 | 1.50 [0.3 to 5.0] | 1.00 [0.3 to 4.0]

2. Secondary Outcome: Cohort 1: Apparent Terminal Phase Half-life (t1/2)
Description: Blood samples were collected for the analysis of PK parameters.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hour (h)
Arm/Group | Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) | Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference)
Number analyzed (Participants) | 30 | 30
Hour (h)
  Day 1: number analyzed (Participants) | 16 | 14
  Day 1 | 7.83 (1.093) | 7.50 (1.731)
  Day 4: number analyzed (Participants) | 14 | 16
  Day 4 | 7.62 (0.904) | 7.43 (1.546)
  Day 7: number analyzed (Participants) | 13 | 15
  Day 7 | 7.92 (2.257) | 7.35 (1.388)
  Day 10: number analyzed (Participants) | 14 | 13
  Day 10 | 8.17 (1.377) | 7.22 (1.319)

3. Secondary Outcome: Cohort 1: Area Under the Plasma Concentration-time Curve up to Last Time With Concentrations Above the Lower Limit of Quantification (LLOQ) (AUC[0-last])
Description: Blood samples were collected for the analysis of PK parameters.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: h*pg/mL
Groups:
- Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test): Healthy participants in cohort 1 received Salbutamol HFA-152a (Test) via MDI as single dose of 200 ug (2 x 100 µg) as inhalation suspension at 20 second intervals on Day 1, Day 4, Day 7 and Day 10.
- Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference): Healthy participants in cohort 1 received Salbutamol HFA-134a (Reference) via MDI as single dose of 200 ug (2 x 100 ug) as inhalation suspension at 20 second intervals on Day 1, Day 4, Day 7 and Day 10
Arm/Group | Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) | Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference)
Number analyzed (Participants) | 30 | 30
h*pg/mL | 5120.73 [4644.42 to 5645.89] | 3977.02 [3674.43 to 4304.54]

4. Secondary Outcome: Cohort 1-Intra-Participant Variability of AUC (0-30min)
Description: Blood samples were collected for the analysis of PK parameters.
Time Frame: At pre-dose, 3, 5, 10, 15, 20 and 30 minutes post-dose on Day 1 (Period 1), Day 4 (Period 2), Day 7 (Period 3) and Day 10 (Period 4)
Population: Pharmacokinetic Population. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field.
Measure: Number; unit: Percentage of Coefficient Variation
Arm/Group | Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) | Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference)
Number analyzed (Participants) | 29 | 29
Percentage of Coefficient Variation | 36.3 | 28.7

5. Secondary Outcome: Cohort 1: Intra Participant Variability of AUC (0-infinity)
Description: Blood samples were collected for the analysis of PK parameters.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Number; unit: Percentage of Coefficient Variation
Arm/Group | Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) | Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference)
Number analyzed (Participants) | 30 | 30
Percentage of Coefficient Variation | 28.3 | 18.6

6. Secondary Outcome: Cohort 1: Intra Participant Variability of AUC(0-last)
Description: Blood samples were collected for the analysis of PK parameters.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Number; unit: Percentage of Coefficient Variation
Arm/Group | Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) | Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference)
Number analyzed (Participants) | 30 | 30
Percentage of Coefficient Variation | 28.5 | 18.3

7. Secondary Outcome: Cohort 1: Intra Participant Variability of Cmax
Description: Blood samples were collected for the analysis of PK parameters.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Number; unit: Percentage of Coefficient Variation
Arm/Group | Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) | Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference)
Number analyzed (Participants) | 30 | 30
Percentage of Coefficient Variation | 33.5 | 17.3

8. Secondary Outcome: Cohort 1: Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose, results in death; was life threatening; required hospitalization or prolongation of existing hospitalization; resulted in disability/incapacity; was a congenital anomaly/birth defect, abnormal pregnancy outcomes. SAEs are subset of AEs. AEs were coded using the Medical Dictionary for Regulatory Activities (MedDRA) coding system.
Time Frame: Up to 46 days [From ICF signing (Day -28) until telephonic follow-up (Day 18)]
Population: Safety Population included all participants who received at least one puff/actuation of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Salbutamol HFA-134a MDI 200 µg (Reference): Healthy participants in cohort 1 received Salbutamol HFA-134a (Reference) via MDI as single dose of 200 ug as inhalation suspension at 20 second intervals administered on Day 4 and Day 7 in the first sequence (TRRT) and Day 1 and Day 10 in the second sequence (RTTR), where R is salbutamol HFA-134a (reference) and T is salbutamol HFA-152a (test).
Arm/Group | Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) | Cohort 1: Salbutamol HFA-134a MDI 200 µg (Reference)
Number analyzed (Participants) | 30 | 30
Participants
  Any AE | 18 | 12
  Any SAE | 1 | 0

9. Secondary Outcome: Cohort 1: Absolute Values for 12 Lead Electrocardiogram (ECGs) Recording of Heart Rate (HR)
Description: A standard 12 lead ECG was obtained using an ECG machine that automatically calculated the HR and were measured after resting for at least 5 minutes in the supine position.
Time Frame: Baseline (pre-dose) and post-dose at 30 minutes on Day 1 [Period 1], Day 4 [Period 2], Day 7 [Period 3], Day 10 [Period 4] and Day 11 (Discharge)
Population: Safety Population. "Overall Number of Participants Analyzed" included the total number of participants in Cohort 1. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) | Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference)
Number analyzed (Participants) | 30 | 30
Beats per minute
  Baseline (Pre-dose at Day 1 [Period 1]): number analyzed (Participants) | 16 | 14
  Baseline (Pre-dose at Day 1 [Period 1]) | 55.1 (6.25) | 52.7 (5.14)
  Post-dose at 30 minutes on Day 1 [Period 1]: number analyzed (Participants) | 16 | 14
  Post-dose at 30 minutes on Day 1 [Period 1] | 63.1 (7.02) | 62.6 (7.56)
  Baseline (Pre-dose at Day 4 [Period 2]): number analyzed (Participants) | 14 | 16
  Baseline (Pre-dose at Day 4 [Period 2]) | 53.6 (6.32) | 55.0 (8.06)
  Post-dose at 30 minutes on Day 4 [Period 2]: number analyzed (Participants) | 14 | 16
  Post-dose at 30 minutes on Day 4 [Period 2] | 62.3 (5.98) | 62.8 (5.75)
  Baseline (Pre-dose at Day 7 [Period 3]): number analyzed (Participants) | 14 | 16
  Baseline (Pre-dose at Day 7 [Period 3]) | 55.4 (7.37) | 56.6 (6.71)
  Post-dose at 30 minutes on Day 7 [Period 3]: number analyzed (Participants) | 14 | 16
  Post-dose at 30 minutes on Day 7 [Period 3] | 67.9 (9.79) | 62.3 (8.68)
  Baseline (Pre-dose at Day 10 [Period 4]): number analyzed (Participants) | 15 | 13
  Baseline (Pre-dose at Day 10 [Period 4]) | 56.5 (6.88) | 53.7 (5.03)
  Post-dose at 30 minutes on Day 10 [Period 4]: number analyzed (Participants) | 15 | 13
  Post-dose at 30 minutes on Day 10 [Period 4] | 64.9 (9.31) | 64.2 (7.83)
  Day 11 (Discharge): number analyzed (Participants) | 15 | 13
  Day 11 (Discharge) | 60.7 (10.59) | 61.2 (8.96)

10. Secondary Outcome: Cohort 1: Absolute Values for 12 Lead ECGs Recording of QT Interval Corrected Using Fridericia's Formula (QTcF) Intervals
Description: A standard 12 lead ECG was obtained using an ECG machine that automatically calculated the QTcF Interval and were measured after resting for at least 5 minutes in the supine position.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) | Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference)
Number analyzed (Participants) | 30 | 30
milliseconds (ms)
  Baseline (Pre-dose at Day 1 [Period 1]): number analyzed (Participants) | 16 | 14
  Baseline (Pre-dose at Day 1 [Period 1]) | 403.0 (16.12) | 411.6 (18.70)
  Post-dose at 30 minutes on Day 1 [Period 1]: number analyzed (Participants) | 16 | 14
  Post-dose at 30 minutes on Day 1 [Period 1] | 396.4 (15.50) | 402.4 (16.22)
  Baseline (Pre-dose at Day 4 [Period 2]): number analyzed (Participants) | 14 | 16
  Baseline (Pre-dose at Day 4 [Period 2]) | 411.9 (18.94) | 399.0 (15.77)
  Post-dose at 30 minutes on Day 4 [Period 2]: number analyzed (Participants) | 14 | 16
  Post-dose at 30 minutes on Day 4 [Period 2] | 400.4 (19.25) | 393.1 (16.80)
  Baseline (Pre-dose at Day 7 [Period 3]): number analyzed (Participants) | 14 | 16
  Baseline (Pre-dose at Day 7 [Period 3]) | 412.4 (18.30) | 397.4 (13.64)
  Post-dose at 30 minutes on Day 7 [Period 3]: number analyzed (Participants) | 14 | 16
  Post-dose at 30 minutes on Day 7 [Period 3] | 403.6 (19.66) | 389.9 (12.09)
  Baseline (Pre-dose at Day 10 [Period 4]): number analyzed (Participants) | 15 | 13
  Baseline (Pre-dose at Day 10 [Period 4]) | 397.6 (13.14) | 411.1 (18.06)
  Post-dose at 30 minutes on Day 10 [Period 4]: number analyzed (Participants) | 15 | 13
  Post-dose at 30 minutes on Day 10 [Period 4] | 392.7 (13.92) | 399.8 (21.48)
  Day 11(Discharge): number analyzed (Participants) | 15 | 13
  Day 11(Discharge) | 388.9 (14.24) | 402.5 (19.75)

11. Secondary Outcome: Cohort 1: Change From Baseline (CFB) for Post-dose 12 Lead ECGs Recording of HR
Description: A standard 12 lead ECG was obtained using an ECG machine that automatically calculated HR and were measured after resting for at least 5 minutes in the supine position.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) | Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference)
Number analyzed (Participants) | 30 | 30
Beats per minute
  CFB to Post-dose at 30 minutes on Day 1 [Period 1]: number analyzed (Participants) | 16 | 14
  CFB to Post-dose at 30 minutes on Day 1 [Period 1] | 8.0 (4.03) | 10.0 (3.84)
  CFB to Post-dose at 30 minutes on Day 4 [Period 2]: number analyzed (Participants) | 14 | 16
  CFB to Post-dose at 30 minutes on Day 4 [Period 2] | 8.6 (3.4) | 7.8 (6.43)
  CFB to Post-dose at 30 minutes on Day 7 [Period 3]: number analyzed (Participants) | 14 | 16
  CFB to Post-dose at 30 minutes on Day 7 [Period 3] | 12.5 (7.62) | 5.7 (4.84)
  CFB to Post-dose at 30 minutes on Day 10 [Period 4]: number analyzed (Participants) | 15 | 13
  CFB to Post-dose at 30 minutes on Day 10 [Period 4] | 8.3 (5.74) | 10.4 (4.79)
  CFB to Day 11 (Discharge): number analyzed (Participants) | 15 | 13
  CFB to Day 11 (Discharge) | 4.1 (7.25) | 7.5 (6.69)

12. Secondary Outcome: Cohort 1: Change From Baseline (CFB) for Post-dose 12 Lead ECGs Recording of QTcF Intervals
Description: as for outcome 10
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) | Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference)
Number analyzed (Participants) | 30 | 30
milliseconds (ms)
  CFB to Post-dose at 30 minutes on Day 1 [Period 1]: number analyzed (Participants) | 16 | 14
  CFB to Post-dose at 30 minutes on Day 1 [Period 1] | -6.6 (12.78) | -9.2 (6.89)
  CFB to Post-dose at 30 minutes on Day 4 [Period 2]: number analyzed (Participants) | 14 | 16
  CFB to Post-dose at 30 minutes on Day 4 [Period 2] | -11.5 (4.83) | -5.9 (13.26)
  CFB to Post-dose at 30 minutes on Day 7 [Period 3]: number analyzed (Participants) | 14 | 16
  CFB to Post-dose at 30 minutes on Day 7 [Period 3] | -8.9 (8.69) | -7.5 (9.04)
  CFB to Post-dose at 30 minutes on Day 10 [Period 4]: number analyzed (Participants) | 15 | 13
  CFB to Post-dose at 30 minutes on Day 10 [Period 4] | -4.9 (12.68) | -11.3 (8.52)
  CFB to Day 11 (Discharge): number analyzed (Participants) | 15 | 13
  CFB to Day 11 (Discharge) | -8.7 (9.29) | -8.5 (9.99)

13. Secondary Outcome: Cohort 1: Absolute Values of Hematology Parameters: Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils and Platelet Count
Description: Blood samples were collected for analyzing absolute values of Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils and Platelet count. Baseline is defined as the latest non-missing pre-dose value
Time Frame: Baseline (Day -1) and Day 11 (Discharge)
Population: Safety Population. As outlined in the protocol, clinical laboratory data were collected at baseline and discharge, hence the data were analyzed and presented by treatment sequence. Each participant was counted only once for this analysis.
Measure: Mean (Standard Deviation); unit: Giga cells/Liter
Arm/Group | Cohort 1: TRRT1 | Cohort 1: RTTR1
Number analyzed (Participants) | 15 | 13
Giga cells/Liter
  Neutrophils: Baseline (Day -1) | 3.62 (1.058) | 3.32 (1.271)
  Neutrophils: Day 11 (Discharge) | 3.05 (0.829) | 2.95 (0.918)
  Lymphocytes: Baseline (Day -1) | 2.07 (0.437) | 1.97 (0.654)
  Lymphocytes: Day 11 (Discharge) | 2.08 (0.707) | 1.88 (0.472)
  Monocytes: Baseline (Day -1) | 0.33 (0.062) | 0.33 (0.075)
  Monocytes: Day 11 (Discharge) | 0.28 (0.094) | 0.32 (0.080)
  Eosinophils: Baseline (Day -1) | 0.13 (0.046) | 0.16 (0.077)
  Eosinophils: Day 11 (Discharge) | 0.11 (0.035) | 0.15 (0.052)
  Basophils: Baseline (Day -1) | 0.03 (0.049) | 0.05 (0.052)
  Basophils: Day 11 (Discharge) | 0.03 (0.049) | 0.03 (0.048)
  Platelet count: Baseline (Day -1) | 254.9 (45.61) | 262.8 (63.27)
  Platelet count: Day 11 (Discharge) | 252.1 (40.26) | 230.6 (50.04)

14. Secondary Outcome: Cohort 1: Absolute Values of Hematology Parameter: Erythrocytes
Description: Blood samples were collected for analyzing absolute values of Erythrocytes. Baseline is defined as the latest non-missing pre-dose value
Time Frame: Baseline (Day -1) and Day 11 (Discharge)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Trillion cells/Liter
Arm/Group | Cohort 1: TRRT1 | Cohort 1: RTTR1
Number analyzed (Participants) | 15 | 13
Trillion cells/Liter
  Baseline (Day -1) | 4.890 (0.4431) | 5.158 (0.4141)
  Day 11 (Discharge) | 4.516 (0.4710) | 4.753 (0.4655)

15. Secondary Outcome: Cohort 1: Absolute Values of Hematology Parameter: Mean Corpuscular Volume (MCV)
Description: Blood samples were collected for analyzing absolute values of Mean Corpuscular Volume (MCV). Baseline is defined as the latest non-missing pre-dose value
Time Frame: Baseline (Day -1) and Day 11 (Discharge)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: femtoliter (fL)
Arm/Group | Cohort 1: TRRT1 | Cohort 1: RTTR1
Number analyzed (Participants) | 15 | 13
femtoliter (fL)
  Baseline (Day -1) | 91.1 (4.61) | 92.1 (3.04)
  Day 11 (Discharge) | 90.0 (4.26) | 91.6 (2.50)

16. Secondary Outcome: Cohort 1: Absolute Values of Hematology Parameter: Mean Corpuscular Hemoglobin (MCH)
Description: Blood samples were collected for analyzing absolute values of Mean corpuscular hemoglobin (MCH). Baseline is defined as the latest non-missing pre-dose value
Time Frame: Baseline (Day -1) and Day 11 (Discharge)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: femtomole (fmol)
Arm/Group | Cohort 1: TRRT1 | Cohort 1: RTTR1
Number analyzed (Participants) | 15 | 13
femtomole (fmol)
  Baseline (Day -1) | 1.817 (0.0977) | 1.845 (0.0599)
  Day 11 (Discharge) | 1.823 (0.1077) | 1.841 (0.0640)

17. Secondary Outcome: Cohort 1: Absolute Values of Hematology Parameter: Hemoglobin
Description: Blood samples were collected for analyzing absolute values of Hemoglobin. Baseline is defined as the latest non-missing pre-dose value
Time Frame: Baseline (Day -1) and Day 11 (Discharge)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Cohort 1: TRRT1 | Cohort 1: RTTR1
Number analyzed (Participants) | 15 | 13
gram per liter (g/L)
  Baseline (Day -1) | 143.19 (14.903) | 153.08 (11.699)
  Day 11 (Discharge) | 132.77 (14.593) | 140.94 (12.026)

18. Secondary Outcome: Cohort 1: Absolute Values of Hematology Parameter: Hematocrit
Description: Blood samples were collected for analyzing absolute values of Hematocrit. Baseline is defined as the latest non-missing pre-dose value
Time Frame: Baseline (Day -1) and Day 11 (Discharge)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Cohort 1: TRRT1 | Cohort 1: RTTR1
Number analyzed (Participants) | 15 | 13
Percentage of red blood cells in blood
  Baseline (Day -1) | 0.445 (0.0405) | 0.475 (0.0355)
  Day 11 (Discharge) | 0.405 (0.0426) | 0.433 (0.0392)

19. Secondary Outcome: Cohort 1: Absolute Values of Clinical Chemistry Parameters, Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST) and Creatine Phosphokinase (CPK)
Description: Blood samples were collected for analyzing absolute values of Alanine aminotransferase (ALT), Alkaline phosphatase (ALP), Aspartate aminotransferase (AST) and Creatine Phosphokinase (CPK). Baseline is defined as the latest non-missing pre-dose value
Time Frame: Baseline (Day -1) and Day 11 (Discharge)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: International Units per Liter (IU/L)
Arm/Group | Cohort 1: TRRT1 | Cohort 1: RTTR1
Number analyzed (Participants) | 15 | 13
International Units per Liter (IU/L)
  ALT: Baseline (Day -1) | 21.67 (9.108) | 23.22 (10.178)
  ALT: Day 11 (Discharge) | 19.33 (5.327) | 21.45 (8.102)
  ALP: Baseline (Day -1) | 65.4 (14.26) | 73.1 (17.89)
  ALP: Day 11 (Discharge) | 60.5 (15.85) | 64.4 (12.41)
  AST: Baseline (Day -1) | 12.38 (3.984) | 14.52 (5.611)
  AST: Day 11 (Discharge) | 10.49 (3.010) | 11.66 (4.240)
  CPK: Baseline (Day -1) | 103.1 (44.25) | 120.4 (60.49)
  CPK: Day 11 (Discharge) | 88.1 (61.28) | 79.9 (32.26)

20. Secondary Outcome: Cohort 1: Absolute Values of Clinical Chemistry Parameters: Direct Bilirubin, Total Bilirubin, Total Protein and Creatinine
Description: Blood samples were collected for analyzing absolute values of direct bilirubin, total bilirubin, total protein and Creatinine. Baseline is defined as the latest non-missing pre-dose value
Time Frame: Baseline (Day -1) and Day 11 (Discharge)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: micromoles per liter (umol/L)
Arm/Group | Cohort 1: TRRT1 | Cohort 1: RTTR1
Number analyzed (Participants) | 15 | 13
micromoles per liter (umol/L)
  Direct Bilirubin: Baseline (Day -1) | 4.12 (2.214) | 4.85 (2.035)
  Direct Bilirubin: Day 11 (Discharge) | 3.79 (2.055) | 4.15 (1.531)
  Total Bilirubin: Baseline (Day -1) | 12.2 (6.22) | 16.3 (7.10)
  Total Bilirubin: Day 11 (Discharge) | 11.8 (5.82) | 13.8 (5.89)
  Total Protein: Baseline (Day -1) | 74.1 (3.75) | 73.3 (4.19)
  Total Protein: Day 11 (Discharge) | 68.2 (3.59) | 66.9 (3.40)
  Creatinine: Baseline (Day -1) | 63.3 (12.48) | 73.6 (18.33)
  Creatinine: Day 11 (Discharge) | 62.1 (10.92) | 69.4 (15.33)

21. Secondary Outcome: Cohort 1: Absolute Values for Chemistry Parameters: Calcium, Sodium, Urea Nitrogen
Description: Blood samples were collected for analyzing absolute values of Calcium, Sodium and Urea Nitrogen. Baseline is defined as the latest non-missing pre-dose value
Time Frame: Baseline (Day -1) and Day 11 (Discharge)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Cohort 1: TRRT1 | Cohort 1: RTTR1
Number analyzed (Participants) | 15 | 13
millimoles per liter (mmol/L)
  Calcium: Baseline (Day -1) | 2.388 (0.0561) | 2.431 (0.0656)
  Calcium: Day 11 (Discharge) | 2.300 (0.0515) | 2.306 (0.0678)
  Sodium: Baseline (Day -1) | 139.7 (2.31) | 139.7 (1.38)
  Sodium: Day 11 (Discharge) | 139.7 (0.90) | 140.3 (1.03)
  Urea Nitrogen: Baseline (Day -1) | 4.12 (0.945) | 4.54 (1.149)
  Urea Nitrogen: Day 11 (Discharge) | 4.28 (0.837) | 4.17 (0.832)

22. Secondary Outcome: Cohort 1: Absolute Values for Chemistry Parameter: Glucose and Potassium
Description: Blood samples were collected for analyzing absolute values of glucose and potassium
Time Frame: Baseline (Pre-dose) and Post-dose at 15, 30 minutes and 1, 1.5, 2 and 4 hours on Day 1 [Period 1], Day 4 [Period 2], Day 7 [Period 3] and Day 10 [ Period 4]
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) | Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference)
Number analyzed (Participants) | 30 | 30
millimoles per liter (mmol/L)
  Baseline (Pre-dose at Day 1 [Period 1]), Glucose: number analyzed (Participants) | 16 | 14
  Baseline (Pre-dose at Day 1 [Period 1]), Glucose | 4.76 (0.206) | 4.89 (0.363)
  Day 1: Post-dose at 15 minutes (Period 1), Glucose: number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 15 minutes (Period 1), Glucose | 4.97 (0.803) | 4.60 (1.060)
  Day 1: Post-dose at 30 minutes (Period 1), Glucose: number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 30 minutes (Period 1), Glucose | 4.86 (0.453) | 4.71 (0.691)
  Day 1: Post-dose at 1 hour (Period 1), Glucose: number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 1 hour (Period 1), Glucose | 5.20 (0.716) | 4.92 (0.415)
  Day 1: Post-dose at 1.5 hours (Period 1), Glucose: number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 1.5 hours (Period 1), Glucose | 4.99 (0.509) | 4.86 (0.271)
  Day 1: Post-dose at 2 hours (Period 1), Glucose: number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 2 hours (Period 1), Glucose | 4.77 (0.322) | 4.72 (0.356)
  Day 1: Post-dose at 4 hours (Period 1), Glucose: number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 4 hours (Period 1), Glucose | 4.50 (0.310) | 4.49 (0.243)
  Baseline (Pre-dose at Day 4 [Period 2]), Glucose: number analyzed (Participants) | 14 | 16
  Baseline (Pre-dose at Day 4 [Period 2]), Glucose | 4.71 (0.284) | 4.65 (0.237)
  Day 4: Post-dose at 15 minutes (Period 2), Glucose: number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 15 minutes (Period 2), Glucose | 4.80 (0.706) | 4.93 (0.758)
  Day 4: Post-dose at 30 minutes (Period 2), Glucose: number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 30 minutes (Period 2), Glucose | 4.70 (0.553) | 4.93 (0.588)
  Day 4: Post-dose at 1 hour (Period 2), Glucose: number analyzed (Participants) | 14 | 15
  Day 4: Post-dose at 1 hour (Period 2), Glucose | 4.84 (0.445) | 4.91 (0.488)
  Day 4: Post-dose at 1.5 hours (Period 2), Glucose: number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 1.5 hours (Period 2), Glucose | 4.74 (0.346) | 4.78 (0.431)
  Day 4: Post-dose at 2 hours (Period 2), Glucose: number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 2 hours (Period 2), Glucose | 4.71 (0.196) | 4.61 (0.427)
  Day 4: Post-dose at 4 hours (Period 2), Glucose: number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 4 hours (Period 2), Glucose | 4.57 (0.258) | 4.53 (0.355)
  Baseline (Pre-dose at Day 7 [Period 3]), Glucose: number analyzed (Participants) | 14 | 16
  Baseline (Pre-dose at Day 7 [Period 3]), Glucose | 4.63 (0.307) | 4.59 (0.232)
  Day 7: Post-dose at 15 minutes (Period 3), Glucose: number analyzed (Participants) | 13 | 16
  Day 7: Post-dose at 15 minutes (Period 3), Glucose | 4.66 (0.852) | 5.02 (0.895)
  Day 7: Post-dose at 30 minutes (Period 3), Glucose: number analyzed (Participants) | 13 | 16
  Day 7: Post-dose at 30 minutes (Period 3), Glucose | 4.56 (0.577) | 4.88 (0.680)
  Day 7: Post-dose at 1 hour (Period 3), Glucose: number analyzed (Participants) | 14 | 16
  Day 7: Post-dose at 1 hour (Period 3), Glucose | 4.75 (0.320) | 4.68 (0.449)
  Day 7: Post-dose at 1.5 hours (Period 3), Glucose: number analyzed (Participants) | 14 | 16
  Day 7: Post-dose at 1.5 hours (Period 3), Glucose | 4.76 (0.414) | 4.72 (0.369)
  Day 7: Post-dose at 2 hours (Period 3), Glucose: number analyzed (Participants) | 14 | 16
  Day 7: Post-dose at 2 hours (Period 3), Glucose | 4.57 (0.358) | 4.49 (0.286)
  Day 7: Post-dose at 4 hours (Period 3), Glucose: number analyzed (Participants) | 13 | 16
  Day 7: Post-dose at 4 hours (Period 3), Glucose | 4.51 (0.236) | 4.51 (0.299)
  Baseline (Pre-dose at Day 10 (Period 4), Glucose: number analyzed (Participants) | 15 | 13
  Baseline (Pre-dose at Day 10 (Period 4), Glucose | 4.62 (0.283) | 4.66 (0.166)
  Day 10: Post-dose at 15 minutes (Period 4), Glucose: number analyzed (Participants) | 15 | 13
  Day 10: Post-dose at 15 minutes (Period 4), Glucose | 4.97 (0.701) | 4.99 (0.856)
  Day 10: Post-dose at 30 minutes (Period 4), Glucose: number analyzed (Participants) | 15 | 13
  Day 10: Post-dose at 30 minutes (Period 4), Glucose | 4.90 (0.650) | 4.98 (0.938)
  Day 10: Post-dose at 1 hour (Period 4), Glucose: number analyzed (Participants) | 14 | 13
  Day 10: Post-dose at 1 hour (Period 4), Glucose | 5.01 (0.476) | 4.92 (0.518)
  Day 10: Post-dose at 1.5 hours (Period 4), Glucose: number analyzed (Participants) | 15 | 12
  Day 10: Post-dose at 1.5 hours (Period 4), Glucose | 4.60 (0.280) | 4.86 (0.548)
  Day 10: Post-dose at 2 hours (Period 4), Glucose: number analyzed (Participants) | 15 | 13
  Day 10: Post-dose at 2 hours (Period 4), Glucose | 4.47 (0.246) | 4.59 (0.278)
  Day 10: Post-dose at 4 hours (Period 4), Glucose: number analyzed (Participants) | 15 | 13
  Day 10: Post-dose at 4 hours (Period 4), Glucose | 4.55 (0.304) | 4.48 (0.239)
  Baseline (Pre-dose at Day 1 [Period 1]), Potassium: number analyzed (Participants) | 16 | 14
  Baseline (Pre-dose at Day 1 [Period 1]), Potassium | 4.19 (0.208) | 4.37 (0.289)
  Day 1: Post-dose at 15 minutes (Period 1), Potassium: number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 15 minutes (Period 1), Potassium | 4.18 (0.261) | 4.29 (0.244)
  Day 1: Post-dose at 30 minutes (Period 1), Potassium: number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 30 minutes (Period 1), Potassium | 4.21 (0.342) | 4.35 (0.241)
  Day 1: Post-dose at 1 hour (Period 1), Potassium: number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 1 hour (Period 1), Potassium | 4.16 (0.175) | 4.24 (0.191)
  Day 1: Post-dose at 1.5 hours (Period 1), Potassium: number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 1.5 hours (Period 1), Potassium | 4.21 (0.188) | 4.49 (0.487)
  Day 1: Post-dose at 2 hours (Period 1), Potassium: number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 2 hours (Period 1), Potassium | 4.20 (0.219) | 4.21 (0.144)
  Day 1: Post-dose at 4 hours (Period 1), Potassium: number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 4 hours (Period 1), Potassium | 4.13 (0.268) | 4.28 (0.255)
  Baseline (Pre-dose at Day 4 [Period 2]), Potassium: number analyzed (Participants) | 14 | 16
  Baseline (Pre-dose at Day 4 [Period 2]), Potassium | 4.33 (0.367) | 4.46 (0.301)
  Day 4: Post-dose at 15 minutes (Period 2), Potassium: number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 15 minutes (Period 2), Potassium | 4.47 (0.307) | 4.21 (0.359)
  Day 4: Post-dose at 30 minutes (Period 2), Potassium: number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 30 minutes (Period 2), Potassium | 4.27 (0.205) | 4.37 (0.793)
  Day 4: Post-dose at 1 hour (Period 2), Potassium: number analyzed (Participants) | 14 | 15
  Day 4: Post-dose at 1 hour (Period 2), Potassium | 4.27 (0.194) | 4.25 (0.264)
  Day 4: Post-dose at 1.5 hours (Period 2), Potassium: number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 1.5 hours (Period 2), Potassium | 4.20 (0.196) | 4.24 (0.175)
  Day 4: Post-dose at 2 hours (Period 2), Potassium: number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 2 hours (Period 2), Potassium | 4.19 (0.188) | 4.24 (0.213)
  Day 4: Post-dose at 4 hours (Period 2), Potassium: number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 4 hours (Period 2), Potassium | 4.12 (0.167) | 4.26 (0.253)
  Baseline (Pre-dose at Day 7 [Period 3]), Potassium: number analyzed (Participants) | 14 | 16
  Baseline (Pre-dose at Day 7 [Period 3]), Potassium | 4.41 (0.337) | 4.35 (0.228)
  Day 7: Post-dose at 15 minutes (Period 3), Potassium: number analyzed (Participants) | 13 | 16
  Day 7: Post-dose at 15 minutes (Period 3), Potassium | 4.18 (0.268) | 4.24 (0.294)
  Day 7: Post-dose at 30 minutes (Period 3), Potassium: number analyzed (Participants) | 13 | 16
  Day 7: Post-dose at 30 minutes (Period 3), Potassium | 4.20 (0.255) | 4.32 (0.256)
  Day 7: Post-dose at 1 hour (Period 3), Potassium: number analyzed (Participants) | 14 | 16
  Day 7: Post-dose at 1 hour (Period 3), Potassium | 4.18 (0.125) | 4.16 (0.163)
  Day 7: Post-dose at 1.5 hours (Period 3), Potassium: number analyzed (Participants) | 14 | 16
  Day 7: Post-dose at 1.5 hours (Period 3), Potassium | 4.26 (0.247) | 4.26 (0.328)
  Day 7: Post-dose at 2 hours (Period 3), Potassium: number analyzed (Participants) | 14 | 16
  Day 7: Post-dose at 2 hours (Period 3), Potassium | 4.12 (0.119) | 4.26 (0.258)
  Day 7: Post-dose at 4 hours (Period 3), Potassium: number analyzed (Participants) | 13 | 16
  Day 7: Post-dose at 4 hours (Period 3), Potassium | 4.12 (0.300) | 4.25 (0.327)
  Baseline (Pre-dose at Day 10 (Period 4), Potassium: number analyzed (Participants) | 15 | 13
  Baseline (Pre-dose at Day 10 (Period 4), Potassium | 4.25 (0.239) | 4.35 (0.282)
  Day 10: Post-dose at 15 minutes (Period 4), Potassium: number analyzed (Participants) | 15 | 13
  Day 10: Post-dose at 15 minutes (Period 4), Potassium | 4.17 (0.167) | 4.16 (0.185)
  Day 10: Post-dose at 30 minutes (Period 4), Potassium: number analyzed (Participants) | 15 | 13
  Day 10: Post-dose at 30 minutes (Period 4), Potassium | 4.21 (0.327) | 4.26 (0.214)
  Day 10: Post-dose at 1 hour (Period 4), Potassium: number analyzed (Participants) | 14 | 13
  Day 10: Post-dose at 1 hour (Period 4), Potassium | 4.22 (0.258) | 4.15 (0.133)
  Day 10: Post-dose at 1.5 hours (Period 4), Potassium: number analyzed (Participants) | 15 | 12
  Day 10: Post-dose at 1.5 hours (Period 4), Potassium | 4.19 (0.233) | 4.13 (0.144)
  Day 10: Post-dose at 2 hours (Period 4), Potassium: number analyzed (Participants) | 15 | 13
  Day 10: Post-dose at 2 hours (Period 4), Potassium | 4.15 (0.200) | 4.13 (0.149)
  Day 10: Post-dose at 4 hours (Period 4), Potassium: number analyzed (Participants) | 15 | 13
  Day 10: Post-dose at 4 hours (Period 4), Potassium | 4.13 (0.167) | 4.12 (0.141)

23. Secondary Outcome: Cohort 1: Absolute Values of Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP measurements were assessed with a completely automated device after the participant has been resting for at least 5 minutes in the supine position. Manual techniques were used only if an automated device was not available.
Time Frame: Baseline (Pre-dose) and Post-dose at 15, 30 minutes and 1, 2 and 4 hours on Day 1 [Period 1], Day 4 [Period 2], Day 7 [Period 3] and Day 10 [ Period 4]
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) | Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference)
Number analyzed (Participants) | 30 | 30
millimeters of mercury (mmHg)
  Baseline (Pre-dose at Day 1 [Period 1]), SBP: number analyzed (Participants) | 16 | 14
  Baseline (Pre-dose at Day 1 [Period 1]), SBP | 108.6 (6.83) | 111.9 (7.24)
  Day 1: Post-dose at 15 minutes (Period 1), SBP: number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 15 minutes (Period 1), SBP | 109.9 (10.19) | 113.9 (4.83)
  Day 1: Post-dose at 30 minutes (Period 1), SBP: number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 30 minutes (Period 1), SBP | 112.2 (8.84) | 115.9 (6.54)
  Day 1: Post-dose at 1 hour (Period 1), SBP: number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 1 hour (Period 1), SBP | 107.9 (11.74) | 112.6 (7.75)
  Day 1: Post-dose at 2 hours (Period 1), SBP: number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 2 hours (Period 1), SBP | 107.9 (9.39) | 107.6 (6.55)
  Day 1: Post-dose at 4 hours (Period 1), SBP: number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 4 hours (Period 1), SBP | 106.8 (9.02) | 109.1 (7.92)
  Baseline (Pre-dose at Day 4 [Period 2]), SBP: number analyzed (Participants) | 14 | 16
  Baseline (Pre-dose at Day 4 [Period 2]), SBP | 110.2 (10.16) | 104.9 (8.99)
  Day 4: Post-dose at 15 minutes (Period 2), SBP: number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 15 minutes (Period 2), SBP | 113.6 (7.52) | 108.3 (8.12)
  Day 4: Post-dose at 30 minutes (Period 2), SBP: number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 30 minutes (Period 2), SBP | 113.9 (7.53) | 112.1 (11.79)
  Day 4: Post-dose at 1 hour (Period 2), SBP: number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 1 hour (Period 2), SBP | 113.0 (9.99) | 107.5 (7.69)
  Day 4: Post-dose at 2 hours (Period 2), SBP: number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 2 hours (Period 2), SBP | 110.4 (11.66) | 104.5 (8.93)
  Day 4: Post-dose at 4 hours (Period 2), SBP: number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 4 hours (Period 2), SBP | 109.3 (9.00) | 104.3 (9.29)
  Baseline (Pre-dose at Day 7 [Period 3]), SBP: number analyzed (Participants) | 14 | 16
  Baseline (Pre-dose at Day 7 [Period 3]), SBP | 110.3 (8.09) | 103.3 (9.75)
  Day 7: Post-dose at 15 minutes (Period 3), SBP: number analyzed (Participants) | 14 | 16
  Day 7: Post-dose at 15 minutes (Period 3), SBP | 111.8 (6.29) | 106.4 (8.63)
  Day 7: Post-dose at 30 minutes (Period 3), SBP: number analyzed (Participants) | 14 | 16
  Day 7: Post-dose at 30 minutes (Period 3), SBP | 116.4 (7.55) | 108.6 (10.65)
  Day 7: Post-dose at 1 hour (Period 3), SBP: number analyzed (Participants) | 14 | 16
  Day 7: Post-dose at 1 hour (Period 3), SBP | 113.2 (7.16) | 104.3 (7.67)
  Day 7: Post-dose at 2 hours (Period 3), SBP: number analyzed (Participants) | 14 | 16
  Day 7: Post-dose at 2 hours (Period 3), SBP | 107.4 (8.38) | 102.4 (9.85)
  Day 7: Post-dose at 4 hours (Period 3), SBP: number analyzed (Participants) | 13 | 16
  Day 7: Post-dose at 4 hours (Period 3), SBP | 110.5 (7.89) | 102.3 (9.26)
  Baseline (Pre-dose at Day 10 (Period 4), SBP: number analyzed (Participants) | 15 | 13
  Baseline (Pre-dose at Day 10 (Period 4), SBP | 108.0 (9.06) | 111.2 (5.20)
  Day 10: Post-dose at 15 minutes (Period 4), SBP: number analyzed (Participants) | 15 | 13
  Day 10: Post-dose at 15 minutes (Period 4), SBP | 107.1 (9.63) | 114.2 (10.43)
  Day 10: Post-dose at 30 minutes (Period 4), SBP: number analyzed (Participants) | 14 | 13
  Day 10: Post-dose at 30 minutes (Period 4), SBP | 109.1 (9.93) | 115.2 (8.41)
  Day 10: Post-dose at 1 hour (Period 4), SBP: number analyzed (Participants) | 14 | 13
  Day 10: Post-dose at 1 hour (Period 4), SBP | 106.7 (10.72) | 112.6 (7.31)
  Day 10: Post-dose at 2 hours (Period 4), SBP: number analyzed (Participants) | 15 | 13
  Day 10: Post-dose at 2 hours (Period 4), SBP | 104.5 (7.36) | 106.1 (7.03)
  Day 10: Post-dose at 4 hours (Period 4), SBP: number analyzed (Participants) | 15 | 13
  Day 10: Post-dose at 4 hours (Period 4), SBP | 105.1 (12.34) | 110.3 (6.45)
  Baseline (Pre-dose at Day 1 [Period 1]), DBP: number analyzed (Participants) | 16 | 14
  Baseline (Pre-dose at Day 1 [Period 1]), DBP | 65.6 (4.47) | 67.8 (6.81)
  Day 1: Post-dose at 15 minutes (Period 1), DBP: number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 15 minutes (Period 1), DBP | 62.7 (6.19) | 66.0 (3.84)
  Day 1: Post-dose at 30 minutes (Period 1), DBP: number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 30 minutes (Period 1), DBP | 65.5 (5.32) | 66.4 (5.02)
  Day 1: Post-dose at 1 hour (Period 1), DBP: number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 1 hour (Period 1), DBP | 62.7 (5.56) | 63.0 (5.66)
  Day 1: Post-dose at 2 hours (Period 1), DBP: number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 2 hours (Period 1), DBP | 63.4 (4.84) | 63.5 (4.90)
  Day 1: Post-dose at 4 hours (Period 1), DBP: number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 4 hours (Period 1), DBP | 63.3 (5.35) | 63.4 (5.29)
  Baseline (Pre-dose at Day 4 [Period 2]), DBP: number analyzed (Participants) | 14 | 16
  Baseline (Pre-dose at Day 4 [Period 2]), DBP | 64.1 (4.24) | 65.3 (5.74)
  Day 4: Post-dose at 15 minutes (Period 2), DBP: number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 15 minutes (Period 2), DBP | 64.9 (4.14) | 63.9 (6.46)
  Day 4: Post-dose at 30 minutes (Period 2), DBP: number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 30 minutes (Period 2), DBP | 63.9 (4.51) | 64.8 (7.33)
  Day 4: Post-dose at 1 hour (Period 2), DBP: number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 1 hour (Period 2), DBP | 62.1 (5.46) | 63.8 (6.38)
  Day 4: Post-dose at 2 hours (Period 2), DBP: number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 2 hours (Period 2), DBP | 63.3 (6.09) | 63.3 (5.99)
  Day 4: Post-dose at 4 hours (Period 2), DBP: number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 4 hours (Period 2), DBP | 61.4 (5.02) | 62.9 (4.24)
  Baseline (Pre-dose at Day 7 [Period 3]), DBP: number analyzed (Participants) | 14 | 16
  Baseline (Pre-dose at Day 7 [Period 3]), DBP | 68.1 (4.91) | 65.0 (4.38)
  Day 7: Post-dose at 15 minutes (Period 3), DBP: number analyzed (Participants) | 14 | 16
  Day 7: Post-dose at 15 minutes (Period 3), DBP | 63.6 (5.53) | 60.7 (5.19)
  Day 7: Post-dose at 30 minutes (Period 3), DBP: number analyzed (Participants) | 14 | 16
  Day 7: Post-dose at 30 minutes (Period 3), DBP | 64.7 (4.91) | 62.3 (4.58)
  Day 7: Post-dose at 1 hour (Period 3), DBP: number analyzed (Participants) | 14 | 16
  Day 7: Post-dose at 1 hour (Period 3), DBP | 64.4 (4.94) | 60.9 (5.14)
  Day 7: Post-dose at 2 hours (Period 3), DBP: number analyzed (Participants) | 14 | 16
  Day 7: Post-dose at 2 hours (Period 3), DBP | 60.7 (5.22) | 62.3 (6.25)
  Day 7: Post-dose at 4 hours (Period 3), DBP: number analyzed (Participants) | 13 | 16
  Day 7: Post-dose at 4 hours (Period 3), DBP | 63.9 (4.75) | 61.6 (7.35)
  Baseline (Pre-dose at Day 10 (Period 4), DBP: number analyzed (Participants) | 15 | 13
  Baseline (Pre-dose at Day 10 (Period 4), DBP | 66.1 (6.46) | 65.1 (3.99)
  Day 10: Post-dose at 15 minutes (Period 4), DBP: number analyzed (Participants) | 15 | 13
  Day 10: Post-dose at 15 minutes (Period 4), DBP | 63.4 (5.44) | 64.6 (6.36)
  Day 10: Post-dose at 30 minutes (Period 4), DBP: number analyzed (Participants) | 14 | 13
  Day 10: Post-dose at 30 minutes (Period 4), DBP | 62.9 (5.19) | 66.5 (6.70)
  Day 10: Post-dose at 1 hour (Period 4), DBP: number analyzed (Participants) | 14 | 13
  Day 10: Post-dose at 1 hour (Period 4), DBP | 63.4 (5.85) | 62.0 (4.16)
  Day 10: Post-dose at 2 hours (Period 4), DBP: number analyzed (Participants) | 15 | 13
  Day 10: Post-dose at 2 hours (Period 4), DBP | 62.5 (5.97) | 62.8 (4.93)
  Day 10: Post-dose at 4 hours (Period 4), DBP: number analyzed (Participants) | 15 | 13
  Day 10: Post-dose at 4 hours (Period 4), DBP | 63.2 (8.79) | 63.0 (3.92)

24. Secondary Outcome: Cohort 1: Absolute Values of Pulse Rate (PR)
Description: Pulse rate measurements were assessed with a completely automated device after the participant has been resting for at least 5 minutes in the supine position. Manual techniques were used only if an automated device was not available.
Time Frame: as for outcome 23
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) | Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference)
Number analyzed (Participants) | 30 | 30
Beats per minute
  Baseline (Pre-dose at Day 1 [Period 1]): number analyzed (Participants) | 16 | 14
  Baseline (Pre-dose at Day 1 [Period 1]) | 55.7 (7.07) | 51.1 (6.27)
  Day 1: Post-dose at 15 minutes (Period 1): number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 15 minutes (Period 1) | 63.9 (8.07) | 65.3 (9.14)
  Day 1: Post-dose at 30 minutes (Period 1): number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 30 minutes (Period 1) | 61.9 (7.02) | 63.6 (10.03)
  Day 1: Post-dose at 1 hour (Period 1): number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 1 hour (Period 1) | 60.0 (7.87) | 58.7 (7.25)
  Day 1: Post-dose at 2 hours (Period 1): number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 2 hours (Period 1) | 57.7 (9.17) | 54.9 (6.79)
  Day 1: Post-dose at 4 hours (Period 1): number analyzed (Participants) | 16 | 14
  Day 1: Post-dose at 4 hours (Period 1) | 55.8 (7.25) | 53.6 (6.25)
  Baseline (Pre-dose at Day 4 [Period 2]): number analyzed (Participants) | 14 | 16
  Baseline (Pre-dose at Day 4 [Period 2]) | 52.7 (7.17) | 54.4 (8.55)
  Day 4: Post-dose at 15 minutes (Period 2): number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 15 minutes (Period 2) | 64.7 (5.31) | 65.3 (6.87)
  Day 4: Post-dose at 30 minutes (Period 2): number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 30 minutes (Period 2) | 62.8 (6.60) | 64.1 (4.44)
  Day 4: Post-dose at 1 hour (Period 2): number analyzed (Participants) | 14 | 15
  Day 4: Post-dose at 1 hour (Period 2) | 62.1 (7.24) | 59.3 (7.11)
  Day 4: Post-dose at 2 hours (Period 2): number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 2 hours (Period 2) | 57.1 (5.20) | 56.8 (8.64)
  Day 4: Post-dose at 4 hours (Period 2): number analyzed (Participants) | 14 | 16
  Day 4: Post-dose at 4 hours (Period 2) | 57.1 (6.41) | 57.9 (10.99)
  Baseline (Pre-dose at Day 7 [Period 3]): number analyzed (Participants) | 14 | 16
  Baseline (Pre-dose at Day 7 [Period 3]) | 54.7 (7.34) | 56.8 (6.01)
  Day 7: Post-dose at 15 minutes (Period 3): number analyzed (Participants) | 14 | 16
  Day 7: Post-dose at 15 minutes (Period 3) | 69.2 (10.98) | 65.6 (9.18)
  Day 7: Post-dose at 30 minutes (Period 3): number analyzed (Participants) | 14 | 16
  Day 7: Post-dose at 30 minutes (Period 3) | 65.3 (7.43) | 62.6 (8.41)
  Day 7: Post-dose at 1 hour (Period 3): number analyzed (Participants) | 14 | 16
  Day 7: Post-dose at 1 hour (Period 3) | 63.6 (7.62) | 61.6 (6.73)
  Day 7: Post-dose at 2 hours (Period 3): number analyzed (Participants) | 14 | 16
  Day 7: Post-dose at 2 hours (Period 3) | 59.0 (5.80) | 57.5 (7.84)
  Day 7: Post-dose at 4 hours (Period 3): number analyzed (Participants) | 13 | 16
  Day 7: Post-dose at 4 hours (Period 3) | 59.8 (5.74) | 57.6 (9.26)
  Baseline (Pre-dose at Day 10 (Period 4): number analyzed (Participants) | 15 | 13
  Baseline (Pre-dose at Day 10 (Period 4) | 55.6 (8.56) | 54.5 (5.61)
  Day 10: Post-dose at 15 minutes (Period 4): number analyzed (Participants) | 15 | 13
  Day 10: Post-dose at 15 minutes (Period 4) | 67.5 (7.24) | 68.0 (9.70)
  Day 10: Post-dose at 30 minutes (Period 4): number analyzed (Participants) | 14 | 13
  Day 10: Post-dose at 30 minutes (Period 4) | 65.3 (9.80) | 63.4 (7.98)
  Day 10: Post-dose at 1 hour (Period 4): number analyzed (Participants) | 14 | 13
  Day 10: Post-dose at 1 hour (Period 4) | 63.7 (7.82) | 62.1 (9.12)
  Day 10: Post-dose at 2 hours (Period 4): number analyzed (Participants) | 15 | 13
  Day 10: Post-dose at 2 hours (Period 4) | 58.1 (6.92) | 58.9 (8.41)
  Day 10: Post-dose at 4 hours (Period 4): number analyzed (Participants) | 15 | 13
  Day 10: Post-dose at 4 hours (Period 4) | 58.6 (7.81) | 56.8 (7.51)

25. Secondary Outcome: Cohort 2: Time to Reach Cmax (Tmax)
Description: Blood samples were collected for the analysis of PK parameters.
Time Frame: At pre-dose, 3, 5, 10, 15, 20, 30, and 45 minutes post-dose and at 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose on Day 1 (Period 1), Day 4 (Period 2), Day 7 [ Period 3] and Day 10 [Period 4]
Population: Pharmacokinetic Population. "Overall Number of Participants Analyzed" included the total number of participants in Cohort 2. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Median (Full Range); unit: Hour
Groups:
- Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test): Healthy participants in cohort 2 received Salbutamol HFA-152a via MDI as single dose of 800 ug as inhalation suspension at 20 second intervals administered on Day 1 and Day 10 in the first sequence (TRRT) and Day 4 and Day 7 in the second sequence (RTTR), where T is salbutamol HFA-152a (test) and R is salbutamol HFA-134a (reference).
- Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference): Healthy participants in cohort 2 received Salbutamol HFA-134a (Reference) via MDI as single dose of 800 ug as inhalation suspension at 20 second intervals administered on Day 4 and Day 7 in the first sequence (TRRT) and Day 1 and Day 10 in the second sequence (RTTR), where R is salbutamol HFA-134a (reference) and T is salbutamol HFA-152a (test).
Arm/Group | Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) | Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference)
Number analyzed (Participants) | 30 | 30
Hour
  Day 1: number analyzed (Participants) | 14 | 16
  Day 1 | 1.50 [0.2 to 4.0] | 1.25 [0.3 to 2.0]
  Day 4: number analyzed (Participants) | 15 | 13
  Day 4 | 1.50 [0.5 to 4.0] | 1.50 [0.3 to 5.0]
  Day 7: number analyzed (Participants) | 16 | 13
  Day 7 | 1.50 [0.2 to 5.0] | 1.50 [0.3 to 4.0]
  Day 10: number analyzed (Participants) | 13 | 16
  Day 10 | 1.50 [0.3 to 6.0] | 1.50 [0.1 to 4.0]

26. Secondary Outcome: Cohort 2: Apparent Terminal Phase Half-life (t1/2)
Description: Blood samples were collected for the analysis of PK parameters.
Time Frame: as for outcome 1
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) | Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference)
Number analyzed (Participants) | 30 | 30
Hour
  Day 1: number analyzed (Participants) | 14 | 16
  Day 1 | 8.56 (1.945) | 7.73 (1.162)
  Day 4: number analyzed (Participants) | 15 | 13
  Day 4 | 7.65 (1.022) | 7.79 (1.380)
  Day 7: number analyzed (Participants) | 16 | 13
  Day 7 | 7.61 (1.247) | 7.57 (1.438)
  Day 10: number analyzed (Participants) | 13 | 16
  Day 10 | 7.87 (1.678) | 7.74 (1.613)

27. Secondary Outcome: Cohort 2: Area Under the Plasma Concentration-time Curve up to Last Time With Concentrations Above the Lower Limit of Quantification (LLOQ) (AUC[0-last])
Description: Blood samples were collected for the analysis of PK parameters.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: h*pg/mL
Groups:
- Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test): Healthy participants in cohort 2 received Salbutamol HFA-152a (Test) via MDI as single dose of 800 ug (8 x 100 µg) as inhalation suspension at 20 second intervals on Day 1, Day 4, Day 7 and Day 10.
- Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference): Healthy participants in cohort 2 received Salbutamol HFA-134a (Reference) via MDI as single dose of 800 ug (8 x 100 ug) as inhalation suspension at 20 second intervals on Day 1, Day 4, Day 7 and Day 10.
Arm/Group | Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) | Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference)
Number analyzed (Participants) | 30 | 29
h*pg/mL | 15345.11 [14137.58 to 16655.78] | 12840.80 [12011.17 to 13727.73]

28. Secondary Outcome: Cohort 2-Intra-Participant Variability of AUC (0-30min)
Description: Blood samples were collected for the analysis of PK parameters.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number; unit: Percentage of Coefficient Variation
Arm/Group | Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) | Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference)
Number analyzed (Participants) | 30 | 29
Percentage of Coefficient Variation | 22.9 | 25.8

29. Secondary Outcome: Cohort 2: Intra Participant Variability of AUC (0-infinity)
Description: Blood samples were collected for the analysis of PK parameters.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Number; unit: Percentage of Coefficient Variation
Arm/Group | Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) | Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference)
Number analyzed (Participants) | 30 | 29
Percentage of Coefficient Variation | 10.0 | 8.6

30. Secondary Outcome: Cohort 2: Intra Participant Variability of AUC (0-last)
Description: Blood samples were collected for the analysis of PK parameters.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Number; unit: Percentage of Coefficient Variation
Arm/Group | Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) | Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference)
Number analyzed (Participants) | 30 | 29
Percentage of Coefficient Variation | 10.4 | 9.0

31. Secondary Outcome: Cohort 2: Intra Participant Variability of Cmax
Description: Blood samples were collected for the analysis of PK parameters.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Number; unit: Percentage of Coefficient Variation
Arm/Group | Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) | Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference)
Number analyzed (Participants) | 30 | 29
Percentage of Coefficient Variation | 14.1 | 12.2

32. Secondary Outcome: Cohort 2: Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: as for outcome 8
Time Frame: Up to 46 days [From ICF signing (Day -28) until telephonic follow-up (Day 18)]
Population: Safety Population included all participants who received at least one puff/actuation of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: Salbutamol HFA-134a MDI 800 µg (Reference): Healthy participants in cohort 2 received Salbutamol HFA-134a (Reference) via MDI as single dose of 800 ug as inhalation suspension at 20 second intervals administered on Day 4 and Day 7 in the first sequence (TRRT) and Day 1 and Day 10 in the second sequence (RTTR), where R is salbutamol HFA-134a (reference) and T is salbutamol HFA-152a (test).
Arm/Group | Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) | Cohort 2: Salbutamol HFA-134a MDI 800 µg (Reference)
Number analyzed (Participants) | 30 | 30
Participants
  Any AE | 20 | 21
  Any SAE | 0 | 0

33. Secondary Outcome: Cohort 2: Absolute Values for 12 Lead Electrocardiogram (ECGs) Recording of Heart Rate (HR)
Description: as for outcome 9
Time Frame: as for outcome 9
Population: Safety Population. "Overall Number of Participants Analyzed" included the total number of participants in Cohort 2. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) | Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference)
Number analyzed (Participants) | 30 | 30
Beats per minute
  Baseline (Pre-dose at Day 1 [Period 1]): number analyzed (Participants) | 14 | 16
  Baseline (Pre-dose at Day 1 [Period 1]) | 63.9 (13.10) | 53.2 (7.91)
  Post-dose at 30 minutes on Day 1 (Period 1): number analyzed (Participants) | 14 | 16
  Post-dose at 30 minutes on Day 1 (Period 1) | 75.9 (14.29) | 66.4 (7.27)
  Baseline (Pre-dose at Day 4 [Period 2]): number analyzed (Participants) | 16 | 14
  Baseline (Pre-dose at Day 4 [Period 2]) | 54.5 (7.76) | 61.4 (9.38)
  Post-dose at 30 minutes on Day 4 (Period 2): number analyzed (Participants) | 16 | 14
  Post-dose at 30 minutes on Day 4 (Period 2) | 66.7 (8.67) | 76.4 (13.83)
  Baseline (Pre-dose at Day 7 [Period 3]): number analyzed (Participants) | 16 | 13
  Baseline (Pre-dose at Day 7 [Period 3]) | 55.1 (8.38) | 64.1 (10.77)
  Post-dose at 30 minutes on Day 7 (Period 3): number analyzed (Participants) | 16 | 13
  Post-dose at 30 minutes on Day 7 (Period 3) | 66.7 (8.65) | 75.2 (10.17)
  Baseline (Pre-dose at Day 10 [Period 4]): number analyzed (Participants) | 13 | 16
  Baseline (Pre-dose at Day 10 [Period 4]) | 64.1 (9.09) | 55.4 (8.04)
  Post-dose at 30 minutes on Day 10 (Period 4): number analyzed (Participants) | 13 | 16
  Post-dose at 30 minutes on Day 10 (Period 4) | 77.1 (11.11) | 68.4 (9.49)
  Day 11 (Discharge): number analyzed (Participants) | 13 | 16
  Day 11 (Discharge) | 67.8 (10.68) | 59.4 (10.65)

34. Secondary Outcome: Cohort 2: Absolute Values for 12 Lead ECGs Recording of QTcF Intervals
Description: as for outcome 10
Time Frame: as for outcome 9
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) | Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference)
Number analyzed (Participants) | 30 | 30
milliseconds (ms)
  Baseline (Pre-dose at Day 1 [Period 1]): number analyzed (Participants) | 14 | 16
  Baseline (Pre-dose at Day 1 [Period 1]) | 407.8 (17.31) | 399.9 (21.05)
  Post-dose at 30 minutes on Day 1 (Period 1): number analyzed (Participants) | 14 | 16
  Post-dose at 30 minutes on Day 1 (Period 1) | 400.8 (17.71) | 402.9 (18.43)
  Baseline (Pre-dose at Day 4 [Period 2]): number analyzed (Participants) | 16 | 14
  Baseline (Pre-dose at Day 4 [Period 2]) | 398.9 (25.14) | 401.9 (17.55)
  Post-dose at 30 minutes on Day 4 (Period 2): number analyzed (Participants) | 16 | 14
  Post-dose at 30 minutes on Day 4 (Period 2) | 399.6 (23.18) | 401.9 (19.28)
  Baseline (Pre-dose at Day 7 [Period 3]): number analyzed (Participants) | 16 | 13
  Baseline (Pre-dose at Day 7 [Period 3]) | 399.9 (24.76) | 402.7 (17.59)
  Post-dose at 30 minutes on Day 7 (Period 3): number analyzed (Participants) | 16 | 13
  Post-dose at 30 minutes on Day 7 (Period 3) | 402.5 (23.59) | 407.8 (24.84)
  Baseline (Pre-dose at Day 10 [Period 4]): number analyzed (Participants) | 13 | 16
  Baseline (Pre-dose at Day 10 [Period 4]) | 401.8 (15.07) | 397.7 (22.86)
  Post-dose at 30 minutes on Day 10 (Period 4): number analyzed (Participants) | 13 | 16
  Post-dose at 30 minutes on Day 10 (Period 4) | 400.2 (12.76) | 400.6 (22.53)
  Day 11 (Discharge): number analyzed (Participants) | 13 | 16
  Day 11 (Discharge) | 395.9 (18.19) | 391.2 (22.25)

35. Secondary Outcome: Cohort 2: Change From Baseline (CFB) for Post-dose 12 Lead ECGs Recording of HR
Description: as for outcome 11
Time Frame: as for outcome 9
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) | Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference)
Number analyzed (Participants) | 30 | 30
Beats per minute
  CFB to Post-dose at 30 minutes on Day 1 [Period 1]: number analyzed (Participants) | 14 | 16
  CFB to Post-dose at 30 minutes on Day 1 [Period 1] | 12.0 (8.45) | 13.2 (4.51)
  CFB to Post-dose at 30 minutes on Day 4 [Period 2]: number analyzed (Participants) | 16 | 14
  CFB to Post-dose at 30 minutes on Day 4 [Period 2] | 12.2 (4.99) | 15.0 (9.10)
  CFB to Post-dose at 30 minutes on Day 7 [Period 3]: number analyzed (Participants) | 16 | 13
  CFB to Post-dose at 30 minutes on Day 7 [Period 3] | 11.6 (4.52) | 11.1 (4.51)
  CFB to Post-dose at 30 minutes on Day 10 [Period 4]: number analyzed (Participants) | 13 | 16
  CFB to Post-dose at 30 minutes on Day 10 [Period 4] | 12.9 (7.17) | 13.0 (6.31)
  CFB to Day 11 (Discharge): number analyzed (Participants) | 13 | 16
  CFB to Day 11 (Discharge) | 3.7 (5.21) | 4.0 (4.81)

36. Secondary Outcome: Cohort 2: Change From Baseline (CFB) for Post-dose 12 Lead ECGs Recording of QTcF Intervals
Description: as for outcome 10
Time Frame: as for outcome 9
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) | Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference)
Number analyzed (Participants) | 30 | 30
milliseconds
  CFB to Post-dose at 30 minutes on Day 1 [Period 1]: number analyzed (Participants) | 14 | 16
  CFB to Post-dose at 30 minutes on Day 1 [Period 1] | -7.0 (6.96) | 3.0 (10.59)
  CFB to Post-dose at 30 minutes on Day 4 [Period 2]: number analyzed (Participants) | 16 | 14
  CFB to Post-dose at 30 minutes on Day 4 [Period 2] | 0.7 (9.87) | 0.0 (14.23)
  CFB to Post-dose at 30 minutes on Day 7 [Period 3]: number analyzed (Participants) | 16 | 13
  CFB to Post-dose at 30 minutes on Day 7 [Period 3] | 2.6 (11.18) | 5.1 (16.88)
  CFB to Post-dose at 30 minutes on Day 10 [Period 4]: number analyzed (Participants) | 13 | 16
  CFB to Post-dose at 30 minutes on Day 10 [Period 4] | -1.7 (5.52) | 2.9 (8.88)
  CFB to Day 11 (Discharge): number analyzed (Participants) | 13 | 16
  CFB to Day 11 (Discharge) | -5.9 (9.40) | -6.5 (8.79)

37. Secondary Outcome: Cohort 2: Absolute Values of Hematology Parameters: Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils and Platelet Count
Description: as for outcome 13
Time Frame: Baseline (Day -1) and Day 11 (Discharge)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Giga cells/Liter
Arm/Group | Cohort 2: TRRT2 | Cohort 2: RTTR2
Number analyzed (Participants) | 13 | 16
Giga cells/Liter
  Neutrophils: Baseline (Day -1) | 4.56 (1.563) | 3.11 (0.559)
  Neutrophils: Day 11 (Discharge) | 4.20 (1.344) | 2.81 (0.521)
  Lymphocytes: Baseline (Day -1) | 2.17 (0.397) | 2.01 (0.359)
  Lymphocytes: Day 11 (Discharge) | 2.05 (0.431) | 1.98 (0.340)
  Monocytes: Baseline (Day -1) | 0.35 (0.113) | 0.34 (0.089)
  Monocytes: Day 11 (Discharge) | 0.34 (0.096) | 0.33 (0.095)
  Eosinophils: Baseline (Day -1) | 0.12 (0.044) | 0.13 (0.060)
  Eosinophils: Day 11 (Discharge) | 0.15 (0.052) | 0.16 (0.150)
  Basophils: Baseline (Day -1) | 0.03 (0.048) | 0.02 (0.040)
  Basophils: Day 11 (Discharge) | 0.00 (0.000) | 0.01 (0.025)
  Platelet count: Baseline (Day -1) | 276.1 (49.55) | 219.3 (46.78)
  Platelet count: Day 11 (Discharge) | 280.5 (67.17) | 221.3 (53.04)

38. Secondary Outcome: Cohort 2: Absolute Values of Hematology Parameter: Erythrocytes
Description: as for outcome 14
Time Frame: Baseline (Day -1) and Day 11 (Discharge)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Trillion cells/Liter
Arm/Group | Cohort 2: TRRT2 | Cohort 2: RTTR2
Number analyzed (Participants) | 13 | 16
Trillion cells/Liter
  Baseline (Day -1) | 5.028 (0.6223) | 5.038 (0.4072)
  Day 11 (Discharge) | 4.575 (0.5669) | 4.826 (0.4039)

39. Secondary Outcome: Cohort 2: Absolute Values of Hematology Parameter: Mean Corpuscular Volume (MCV)
Description: as for outcome 15
Time Frame: Baseline (Day -1) and Day 11 (Discharge)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: femtoliter (fL)
Arm/Group | Cohort 2: TRRT2 | Cohort 2: RTTR2
Number analyzed (Participants) | 13 | 16
femtoliter (fL)
  Baseline (Day -1) | 89.8 (4.10) | 91.3 (4.51)
  Day 11 (Discharge) | 90.3 (3.99) | 91.4 (4.21)

40. Secondary Outcome: Cohort 2: Absolute Values of Hematology Parameter: Mean Corpuscular Hemoglobin (MCH)
Description: as for outcome 16
Time Frame: Baseline (Day -1) and Day 11 (Discharge)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: femtomole (fmol)
Arm/Group | Cohort 2: TRRT2 | Cohort 2: RTTR2
Number analyzed (Participants) | 13 | 16
femtomole (fmol)
  Baseline (Day -1) | 1.834 (0.0868) | 1.851 (0.0808)
  Day 11 (Discharge) | 1.837 (0.0980) | 1.853 (0.0919)

41. Secondary Outcome: Cohort 2: Absolute Values of Hematology Parameter: Hemoglobin
Description: as for outcome 17
Time Frame: Baseline (Day -1) and Day 11 (Discharge)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Cohort 2: TRRT2 | Cohort 2: RTTR2
Number analyzed (Participants) | 13 | 16
gram per liter (g/L)
  Baseline (Day -1) | 148.25 (18.566) | 149.95 (11.278)
  Day 11 (Discharge) | 134.99 (16.590) | 143.73 (12.170)

42. Secondary Outcome: Cohort 2: Absolute Values of Hematology Parameter: Hematocrit
Description: as for outcome 18
Time Frame: Baseline (Day -1) and Day 11 (Discharge)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Cohort 2: TRRT2 | Cohort 2: RTTR2
Number analyzed (Participants) | 13 | 16
Percentage of red blood cells in blood
  Baseline (Day -1) | 0.450 (0.0537) | 0.458 (0.0338)
  Day 11 (Discharge) | 0.412 (0.0487) | 0.440 (0.0344)

43. Secondary Outcome: Cohort 2: Absolute Values of Clinical Chemistry Parameters, Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST) and Creatine Phosphokinase (CPK)
Description: as for outcome 19
Time Frame: Baseline (Day -1) and Day 11 (Discharge)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: International Units per Liter (IU/L)
Arm/Group | Cohort 2: TRRT2 | Cohort 2: RTTR2
Number analyzed (Participants) | 13 | 16
International Units per Liter (IU/L)
  Baseline (Day -1), ALT | 19.15 (10.383) | 23.88 (11.661)
  Day 11 (Discharge), ALT | 21.22 (9.945) | 25.63 (18.822)
  Baseline (Day -1), ALP | 64.1 (14.94) | 62.6 (22.40)
  Day 11 (Discharge), ALP | 59.8 (12.94) | 60.1 (20.92)
  Baseline (Day -1), AST | 11.13 (3.261) | 14.62 (7.533)
  Day 11 (Discharge), AST | 10.12 (2.481) | 13.72 (13.046)
  Baseline (Day -1), CPK | 87.8 (47.25) | 152.8 (72.50)
  Day 11 (Discharge), CPK | 60.9 (22.91) | 90.0 (34.09)

44. Secondary Outcome: Cohort 2: Absolute Values of Clinical Chemistry Parameters: Direct Bilirubin, Total Bilirubin, Total Protein and Creatinine
Description: as for outcome 20
Time Frame: Baseline (Day -1) and Day 11 (Discharge)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: micromoles per liter (umol/L)
Arm/Group | Cohort 2: TRRT2 | Cohort 2: RTTR2
Number analyzed (Participants) | 13 | 16
micromoles per liter (umol/L)
  Baseline (Day -1), Direct Bilirubin | 3.75 (2.021) | 4.68 (2.537)
  Day 11 (Discharge), Direct Bilirubin | 3.58 (2.523) | 4.18 (2.461)
  Baseline (Day -1), Total Bilirubin | 16.7 (16.45) | 16.1 (9.16)
  Day 11 (Discharge), Total Bilirubin | 11.8 (8.65) | 13.9 (8.43)
  Baseline (Day -1), Total Protein | 74.8 (2.41) | 71.8 (3.69)
  Day 11 (Discharge), Total Protein | 68.0 (3.14) | 68.6 (4.38)
  Baseline (Day -1), Creatinine | 64.8 (12.69) | 71.9 (12.30)
  Day 11 (Discharge), Creatinine | 61.6 (12.91) | 71.4 (12.77)

45. Secondary Outcome: Cohort 2: Absolute Values for Chemistry Parameters: Calcium, Sodium, Urea Nitrogen
Description: as for outcome 21
Time Frame: Baseline (Day -1) and Day 11 (Discharge)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Cohort 2: TRRT2 | Cohort 2: RTTR2
Number analyzed (Participants) | 13 | 16
millimoles per liter (mmol/L)
  Baseline (Day -1), Calcium | 2.422 (0.1248) | 2.388 (0.0683)
  Day 11 (Discharge), Calcium | 2.313 (0.0598) | 2.341 (0.1008)
  Baseline (Day -1), Sodium | 138.8 (1.69) | 139.1 (2.35)
  Day 11 (Discharge), Sodium | 139.8 (1.77) | 140.4 (1.55)
  Baseline (Day -1), Urea Nitrogen | 4.33 (1.637) | 5.39 (0.998)
  Day 11 (Discharge), Urea Nitrogen | 4.18 (0.877) | 4.38 (0.913)

46. Secondary Outcome: Cohort 2: Absolute Values for Chemistry Parameter: Glucose and Potassium
Description: Blood samples were collected for analyzing absolute values of glucose and potassium
Time Frame: as for outcome 22
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) | Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference)
Number analyzed (Participants) | 30 | 30
millimoles per liter (mmol/L)
  Baseline (Pre-dose at Day 1 [Period 1]), Glucose: number analyzed (Participants) | 14 | 16
  Baseline (Pre-dose at Day 1 [Period 1]), Glucose | 4.84 (0.303) | 4.99 (0.336)
  Day 1: Post-dose at 15 minutes (Period 1), Glucose: number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 15 minutes (Period 1), Glucose | 5.04 (0.804) | 4.96 (1.030)
  Day 1: Post-dose at 30 minutes (Period 1), Glucose: number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 30 minutes (Period 1), Glucose | 5.08 (0.558) | 4.96 (0.623)
  Day 1: Post-dose at 1 hour (Period 1), Glucose: number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 1 hour (Period 1), Glucose | 5.26 (0.403) | 4.96 (0.320)
  Day 1: Post-dose at 1.5 hours (Period 1), Glucose: number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 1.5 hours (Period 1), Glucose | 5.09 (0.474) | 4.98 (0.277)
  Day 1: Post-dose at 2 hours (Period 1), Glucose: number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 2 hours (Period 1), Glucose | 4.94 (0.422) | 4.88 (0.349)
  Day 1: Post-dose at 4 hours (Period 1), Glucose: number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 4 hours (Period 1), Glucose | 4.59 (0.297) | 4.74 (0.239)
  Baseline (Pre-dose at Day 4 [Period 2]), Glucose: number analyzed (Participants) | 16 | 14
  Baseline (Pre-dose at Day 4 [Period 2]), Glucose | 4.81 (0.253) | 4.74 (0.334)
  Day 4: Post-dose at 15 minutes (Period 2), Glucose: number analyzed (Participants) | 15 | 13
  Day 4: Post-dose at 15 minutes (Period 2), Glucose | 4.97 (1.605) | 4.72 (0.998)
  Day 4: Post-dose at 30 minutes (Period 2), Glucose: number analyzed (Participants) | 16 | 13
  Day 4: Post-dose at 30 minutes (Period 2), Glucose | 4.89 (1.056) | 4.96 (0.658)
  Day 4: Post-dose at 1 hour (Period 2), Glucose: number analyzed (Participants) | 16 | 13
  Day 4: Post-dose at 1 hour (Period 2), Glucose | 4.88 (0.473) | 4.97 (0.397)
  Day 4: Post-dose at 1.5 hours (Period 2), Glucose: number analyzed (Participants) | 16 | 13
  Day 4: Post-dose at 1.5 hours (Period 2), Glucose | 4.92 (0.550) | 4.78 (0.444)
  Day 4: Post-dose at 2 hours (Period 2), Glucose: number analyzed (Participants) | 16 | 13
  Day 4: Post-dose at 2 hours (Period 2), Glucose | 4.74 (0.334) | 4.54 (0.371)
  Day 4: Post-dose at 4 hours (Period 2), Glucose: number analyzed (Participants) | 16 | 13
  Day 4: Post-dose at 4 hours (Period 2), Glucose | 4.66 (0.225) | 4.52 (0.308)
  Baseline (Pre-dose at Day 7 [Period 3]), Glucose: number analyzed (Participants) | 16 | 13
  Baseline (Pre-dose at Day 7 [Period 3]), Glucose | 4.84 (0.242) | 4.72 (0.368)
  Day 7: Post-dose at 15 minutes (Period 3), Glucose: number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 15 minutes (Period 3), Glucose | 5.01 (0.936) | 5.07 (0.948)
  Day 7: Post-dose at 30 minutes (Period 3), Glucose: number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 30 minutes (Period 3), Glucose | 4.75 (0.516) | 5.05 (0.715)
  Day 7: Post-dose at 1 hour (Period 3), Glucose: number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 1 hour (Period 3), Glucose | 4.84 (0.426) | 5.05 (0.425)
  Day 7: Post-dose at 1.5 hours (Period 3), Glucose: number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 1.5 hours (Period 3), Glucose | 4.73 (0.382) | 5.02 (0.400)
  Day 7: Post-dose at 2 hours (Period 3), Glucose: number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 2 hours (Period 3), Glucose | 4.66 (0.359) | 4.68 (0.383)
  Day 7: Post-dose at 4 hours (Period 3), Glucose: number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 4 hours (Period 3), Glucose | 4.71 (0.154) | 4.57 (0.315)
  Baseline (Pre-dose at Day 10 (Period 4), Glucose: number analyzed (Participants) | 13 | 16
  Baseline (Pre-dose at Day 10 (Period 4), Glucose | 4.67 (0.293) | 4.83 (0.286)
  Day 10: Post-dose at 15 minutes (Period 4), Glucose: number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 15 minutes (Period 4), Glucose | 4.62 (0.887) | 5.23 (1.006)
  Day 10: Post-dose at 30 minutes (Period 4), Glucose: number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 30 minutes (Period 4), Glucose | 4.77 (0.786) | 4.91 (0.692)
  Day 10: Post-dose at 1 hour (Period 4), Glucose: number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 1 hour (Period 4), Glucose | 4.88 (0.285) | 4.79 (0.512)
  Day 10: Post-dose at 1.5 hours (Period 4), Glucose: number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 1.5 hours (Period 4), Glucose | 4.81 (0.411) | 4.73 (0.368)
  Day 10: Post-dose at 2 hours (Period 4), Glucose: number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 2 hours (Period 4), Glucose | 4.62 (0.349) | 4.66 (0.316)
  Day 10: Post-dose at 4 hours (Period 4), Glucose: number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 4 hours (Period 4), Glucose | 4.59 (0.355) | 4.68 (0.235)
  Baseline (Pre-dose at Day 1 [Period 1]), Potassium: number analyzed (Participants) | 14 | 16
  Baseline (Pre-dose at Day 1 [Period 1]), Potassium | 4.28 (0.212) | 4.39 (0.295)
  Day 1: Post-dose at 15 minutes (Period 1), Potassium: number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 15 minutes (Period 1), Potassium | 4.36 (0.365) | 4.32 (0.128)
  Day 1: Post-dose at 30 minutes (Period 1), Potassium: number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 30 minutes (Period 1), Potassium | 4.25 (0.301) | 4.37 (0.296)
  Day 1: Post-dose at 1 hour (Period 1), Potassium: number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 1 hour (Period 1), Potassium | 4.22 (0.345) | 4.23 (0.140)
  Day 1: Post-dose at 1.5 hours (Period 1), Potassium: number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 1.5 hours (Period 1), Potassium | 4.20 (0.277) | 4.28 (0.402)
  Day 1: Post-dose at 2 hours (Period 1), Potassium: number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 2 hours (Period 1), Potassium | 4.30 (0.499) | 4.16 (0.131)
  Day 1: Post-dose at 4 hours (Period 1), Potassium: number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 4 hours (Period 1), Potassium | 4.12 (0.142) | 4.06 (0.163)
  Baseline (Pre-dose at Day 4 [Period 2]), Potassium: number analyzed (Participants) | 16 | 14
  Baseline (Pre-dose at Day 4 [Period 2]), Potassium | 4.28 (0.191) | 4.29 (0.209)
  Day 4: Post-dose at 15 minutes (Period 2), Potassium: number analyzed (Participants) | 15 | 13
  Day 4: Post-dose at 15 minutes (Period 2), Potassium | 4.37 (0.235) | 4.10 (0.321)
  Day 4: Post-dose at 30 minutes (Period 2), Potassium: number analyzed (Participants) | 16 | 13
  Day 4: Post-dose at 30 minutes (Period 2), Potassium | 4.31 (0.241) | 4.38 (0.561)
  Day 4: Post-dose at 1 hour (Period 2), Potassium: number analyzed (Participants) | 16 | 13
  Day 4: Post-dose at 1 hour (Period 2), Potassium | 4.19 (0.161) | 4.20 (0.238)
  Day 4: Post-dose at 1.5 hours (Period 2), Potassium: number analyzed (Participants) | 16 | 13
  Day 4: Post-dose at 1.5 hours (Period 2), Potassium | 4.11 (0.139) | 4.27 (0.371)
  Day 4: Post-dose at 2 hours (Period 2), Potassium: number analyzed (Participants) | 16 | 13
  Day 4: Post-dose at 2 hours (Period 2), Potassium | 4.25 (0.515) | 4.13 (0.206)
  Day 4: Post-dose at 4 hours (Period 2), Potassium: number analyzed (Participants) | 16 | 13
  Day 4: Post-dose at 4 hours (Period 2), Potassium | 4.14 (0.271) | 4.18 (0.241)
  Baseline (Pre-dose at Day 7 [Period 3]), Potassium: number analyzed (Participants) | 16 | 13
  Baseline (Pre-dose at Day 7 [Period 3]), Potassium | 4.28 (0.142) | 4.30 (0.153)
  Day 7: Post-dose at 15 minutes (Period 3), Potassium: number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 15 minutes (Period 3), Potassium | 4.13 (0.153) | 4.25 (0.185)
  Day 7: Post-dose at 30 minutes (Period 3), Potassium: number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 30 minutes (Period 3), Potassium | 4.21 (0.216) | 4.31 (0.218)
  Day 7: Post-dose at 1 hour (Period 3), Potassium: number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 1 hour (Period 3), Potassium | 4.14 (0.178) | 4.19 (0.278)
  Day 7: Post-dose at 1.5 hours (Period 3), Potassium: number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 1.5 hours (Period 3), Potassium | 4.27 (0.613) | 4.18 (0.244)
  Day 7: Post-dose at 2 hours (Period 3), Potassium: number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 2 hours (Period 3), Potassium | 4.12 (0.180) | 4.28 (0.339)
  Day 7: Post-dose at 4 hours (Period 3), Potassium: number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 4 hours (Period 3), Potassium | 4.12 (0.279) | 4.20 (0.183)
  Baseline (Pre-dose at Day 10 (Period 4), Potassium: number analyzed (Participants) | 13 | 16
  Baseline (Pre-dose at Day 10 (Period 4), Potassium | 4.52 (0.440) | 4.35 (0.234)
  Day 10: Post-dose at 15 minutes (Period 4), Potassium: number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 15 minutes (Period 4), Potassium | 4.22 (0.249) | 4.29 (0.294)
  Day 10: Post-dose at 30 minutes (Period 4), Potassium: number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 30 minutes (Period 4), Potassium | 4.40 (0.422) | 4.26 (0.193)
  Day 10: Post-dose at 1 hour (Period 4), Potassium: number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 1 hour (Period 4), Potassium | 4.22 (0.231) | 4.20 (0.171)
  Day 10: Post-dose at 1.5 hours (Period 4), Potassium: number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 1.5 hours (Period 4), Potassium | 4.17 (0.180) | 4.13 (0.134)
  Day 10: Post-dose at 2 hours (Period 4), Potassium: number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 2 hours (Period 4), Potassium | 4.22 (0.228) | 4.07 (0.162)
  Day 10: Post-dose at 4 hours (Period 4), Potassium: number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 4 hours (Period 4), Potassium | 4.15 (0.194) | 4.12 (0.256)

47. Secondary Outcome: Cohort 2: Absolute Values of Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: as for outcome 23
Time Frame: as for outcome 23
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: millimeters of mercury(mmHg)
Arm/Group | Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) | Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference)
Number analyzed (Participants) | 30 | 30
millimeters of mercury(mmHg)
  Baseline (Pre-dose at Day 1 [Period 1]), SBP: number analyzed (Participants) | 14 | 16
  Baseline (Pre-dose at Day 1 [Period 1]), SBP | 109.9 (8.61) | 108.3 (6.78)
  Day 1: Post-dose at 15 minutes (Period 1), SBP: number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 15 minutes (Period 1), SBP | 114.9 (12.04) | 113.8 (9.52)
  Day 1: Post-dose at 30 minutes (Period 1), SBP: number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 30 minutes (Period 1), SBP | 114.6 (9.50) | 113.8 (8.71)
  Day 1: Post-dose at 1 hour (Period 1), SBP: number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 1 hour (Period 1), SBP | 110.4 (8.25) | 110.8 (9.66)
  Day 1: Post-dose at 2 hours (Period 1), SBP: number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 2 hours (Period 1), SBP | 106.9 (8.09) | 110.4 (11.43)
  Day 1: Post-dose at 4 hours (Period 1), SBP: number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 4 hours (Period 1), SBP | 109.4 (7.37) | 109.1 (7.05)
  Baseline (Pre-dose at Day 4 [Period 2]), SBP: number analyzed (Participants) | 16 | 14
  Baseline (Pre-dose at Day 4 [Period 2]), SBP | 106.9 (10.16) | 106.6 (8.20)
  Day 4: Post-dose at 15 minutes (Period 2), SBP: number analyzed (Participants) | 16 | 14
  Day 4: Post-dose at 15 minutes (Period 2), SBP | 111.7 (10.44) | 115.2 (11.87)
  Day 4: Post-dose at 30 minutes (Period 2), SBP: number analyzed (Participants) | 16 | 14
  Day 4: Post-dose at 30 minutes (Period 2), SBP | 111.3 (11.47) | 116.4 (11.17)
  Day 4: Post-dose at 1 hour (Period 2), SBP: number analyzed (Participants) | 16 | 14
  Day 4: Post-dose at 1 hour (Period 2), SBP | 110.9 (9.21) | 110.6 (9.87)
  Day 4: Post-dose at 2 hours (Period 2), SBP: number analyzed (Participants) | 16 | 13
  Day 4: Post-dose at 2 hours (Period 2), SBP | 105.8 (7.30) | 105.4 (7.95)
  Day 4: Post-dose at 4 hours (Period 2), SBP: number analyzed (Participants) | 16 | 13
  Day 4: Post-dose at 4 hours (Period 2), SBP | 108.8 (9.64) | 109.2 (10.94)
  Baseline (Pre-dose at Day 7 [Period 3]), SBP: number analyzed (Participants) | 16 | 13
  Baseline (Pre-dose at Day 7 [Period 3]), SBP | 109.9 (8.04) | 107.5 (8.03)
  Day 7: Post-dose at 15 minutes (Period 3), SBP: number analyzed (Participants) | 15 | 13
  Day 7: Post-dose at 15 minutes (Period 3), SBP | 112.9 (12.96) | 112.8 (9.89)
  Day 7: Post-dose at 30 minutes (Period 3), SBP: number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 30 minutes (Period 3), SBP | 112.8 (10.05) | 114.1 (8.71)
  Day 7: Post-dose at 1 hour (Period 3), SBP: number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 1 hour (Period 3), SBP | 110.4 (9.05) | 108.4 (9.77)
  Day 7: Post-dose at 2 hours (Period 3), SBP: number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 2 hours (Period 3), SBP | 107.8 (8.63) | 105.7 (7.90)
  Day 7: Post-dose at 4 hours (Period 3), SBP: number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 4 hours (Period 3), SBP | 109.4 (7.44) | 108.8 (8.04)
  Baseline (Pre-dose at Day 10 (Period 4), SBP: number analyzed (Participants) | 13 | 16
  Baseline (Pre-dose at Day 10 (Period 4), SBP | 108.8 (7.06) | 108.4 (10.20)
  Day 10: Post-dose at 15 minutes (Period 4), SBP: number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 15 minutes (Period 4), SBP | 113.5 (12.44) | 113.9 (12.37)
  Day 10: Post-dose at 30 minutes (Period 4), SBP: number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 30 minutes (Period 4), SBP | 110.8 (8.47) | 112.9 (11.75)
  Day 10: Post-dose at 1 hour (Period 4), SBP: number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 1 hour (Period 4), SBP | 110.1 (11.02) | 111.6 (10.18)
  Day 10: Post-dose at 2 hours (Period 4), SBP: number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 2 hours (Period 4), SBP | 105.3 (9.70) | 108.4 (8.34)
  Day 10: Post-dose at 4 hours (Period 4), SBP: number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 4 hours (Period 4), SBP | 106.5 (9.90) | 108.6 (8.02)
  Baseline (Pre-dose at Day 1 [Period 1]), DBP: number analyzed (Participants) | 14 | 16
  Baseline (Pre-dose at Day 1 [Period 1]), DBP | 68.9 (7.00) | 64.9 (3.59)
  Day 1: Post-dose at 15 minutes (Period 1), DBP: number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 15 minutes (Period 1), DBP | 66.2 (7.29) | 62.6 (5.24)
  Day 1: Post-dose at 30 minutes (Period 1), DBP: number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 30 minutes (Period 1), DBP | 69.1 (6.74) | 63.2 (3.82)
  Day 1: Post-dose at 1 hour (Period 1), DBP: number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 1 hour (Period 1), DBP | 69.4 (7.27) | 61.5 (5.18)
  Day 1: Post-dose at 2 hours (Period 1), DBP: number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 2 hours (Period 1), DBP | 67.4 (6.58) | 62.5 (5.25)
  Day 1: Post-dose at 4 hours (Period 1), DBP: number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 4 hours (Period 1), DBP | 67.3 (6.26) | 64.6 (5.78)
  Baseline (Pre-dose at Day 4 [Period 2]), DBP: number analyzed (Participants) | 16 | 14
  Baseline (Pre-dose at Day 4 [Period 2]), DBP | 64.1 (6.56) | 70.1 (7.09)
  Day 4: Post-dose at 15 minutes (Period 2), DBP: number analyzed (Participants) | 16 | 14
  Day 4: Post-dose at 15 minutes (Period 2), DBP | 61.4 (5.33) | 66.5 (7.91)
  Day 4: Post-dose at 30 minutes (Period 2), DBP: number analyzed (Participants) | 16 | 14
  Day 4: Post-dose at 30 minutes (Period 2), DBP | 61.8 (7.11) | 68.9 (8.53)
  Day 4: Post-dose at 1 hour (Period 2), DBP: number analyzed (Participants) | 16 | 14
  Day 4: Post-dose at 1 hour (Period 2), DBP | 61.4 (4.30) | 67.9 (8.11)
  Day 4: Post-dose at 2 hours (Period 2), DBP: number analyzed (Participants) | 16 | 13
  Day 4: Post-dose at 2 hours (Period 2), DBP | 60.9 (4.53) | 66.9 (5.88)
  Day 4: Post-dose at 4 hours (Period 2), DBP: number analyzed (Participants) | 16 | 13
  Day 4: Post-dose at 4 hours (Period 2), DBP | 63.1 (5.44) | 68.5 (7.45)
  Baseline (Pre-dose at Day 7 [Period 3]), DBP: number analyzed (Participants) | 16 | 13
  Baseline (Pre-dose at Day 7 [Period 3]), DBP | 65.8 (5.30) | 70.6 (7.83)
  Day 7: Post-dose at 15 minutes (Period 3), DBP: number analyzed (Participants) | 15 | 13
  Day 7: Post-dose at 15 minutes (Period 3), DBP | 63.0 (4.26) | 67.5 (7.01)
  Day 7: Post-dose at 30 minutes (Period 3), DBP: number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 30 minutes (Period 3), DBP | 63.0 (4.58) | 66.6 (6.50)
  Day 7: Post-dose at 1 hour (Period 3), DBP: number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 1 hour (Period 3), DBP | 62.7 (3.48) | 65.8 (7.96)
  Day 7: Post-dose at 2 hours (Period 3), DBP: number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 2 hours (Period 3), DBP | 62.9 (3.92) | 67.0 (5.12)
  Day 7: Post-dose at 4 hours (Period 3), DBP: number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 4 hours (Period 3), DBP | 64.4 (4.73) | 68.5 (7.48)
  Baseline (Pre-dose at Day 10 (Period 4), DBP: number analyzed (Participants) | 13 | 16
  Baseline (Pre-dose at Day 10 (Period 4), DBP | 67.6 (6.76) | 64.9 (4.94)
  Day 10: Post-dose at 15 minutes (Period 4), DBP: number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 15 minutes (Period 4), DBP | 67.8 (7.78) | 62.2 (6.75)
  Day 10: Post-dose at 30 minutes (Period 4), DBP: number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 30 minutes (Period 4), DBP | 67.0 (6.92) | 61.1 (6.77)
  Day 10: Post-dose at 1 hour (Period 4), DBP: number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 1 hour (Period 4), DBP | 66.8 (7.83) | 62.8 (5.21)
  Day 10: Post-dose at 2 hours (Period 4), DBP: number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 2 hours (Period 4), DBP | 66.2 (6.62) | 62.5 (5.30)
  Day 10: Post-dose at 4 hours (Period 4), DBP: number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 4 hours (Period 4), DBP | 66.0 (7.97) | 61.1 (4.40)

48. Secondary Outcome: Cohort 2: Absolute Values of Pulse Rate (PR)
Description: as for outcome 24
Time Frame: as for outcome 23
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) | Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference)
Number analyzed (Participants) | 30 | 30
Beats per minute
  Baseline (Pre-dose at Day 1 [Period 1]): number analyzed (Participants) | 14 | 16
  Baseline (Pre-dose at Day 1 [Period 1]) | 62.1 (11.55) | 51.3 (8.75)
  Day 1: Post-dose at 15 minutes (Period 1): number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 15 minutes (Period 1) | 75.8 (13.49) | 67.7 (8.24)
  Day 1: Post-dose at 30 minutes (Period 1): number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 30 minutes (Period 1) | 75.8 (14.89) | 64.0 (9.15)
  Day 1: Post-dose at 1 hour (Period 1): number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 1 hour (Period 1) | 73.0 (18.02) | 61.1 (8.30)
  Day 1: Post-dose at 2 hours (Period 1): number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 2 hours (Period 1) | 69.8 (13.26) | 57.4 (8.33)
  Day 1: Post-dose at 4 hours (Period 1): number analyzed (Participants) | 14 | 16
  Day 1: Post-dose at 4 hours (Period 1) | 66.6 (14.31) | 56.4 (8.38)
  Baseline (Pre-dose at Day 4 [Period 2]): number analyzed (Participants) | 16 | 14
  Baseline (Pre-dose at Day 4 [Period 2]) | 56.4 (5.90) | 62.1 (10.92)
  Day 4: Post-dose at 15 minutes (Period 2): number analyzed (Participants) | 16 | 14
  Day 4: Post-dose at 15 minutes (Period 2) | 67.1 (7.22) | 77.6 (14.54)
  Day 4: Post-dose at 30 minutes (Period 2): number analyzed (Participants) | 16 | 14
  Day 4: Post-dose at 30 minutes (Period 2) | 64.8 (8.12) | 74.8 (14.48)
  Day 4: Post-dose at 1 hour (Period 2): number analyzed (Participants) | 16 | 14
  Day 4: Post-dose at 1 hour (Period 2) | 64.3 (8.27) | 72.9 (11.04)
  Day 4: Post-dose at 2 hours (Period 2): number analyzed (Participants) | 16 | 13
  Day 4: Post-dose at 2 hours (Period 2) | 60.0 (6.29) | 67.1 (11.27)
  Day 4: Post-dose at 4 hours (Period 2): number analyzed (Participants) | 16 | 13
  Day 4: Post-dose at 4 hours (Period 2) | 57.3 (7.50) | 63.9 (9.84)
  Baseline (Pre-dose at Day 7 [Period 3]): number analyzed (Participants) | 16 | 13
  Baseline (Pre-dose at Day 7 [Period 3]) | 54.9 (8.29) | 64.3 (11.12)
  Day 7: Post-dose at 15 minutes (Period 3): number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 15 minutes (Period 3) | 68.8 (7.93) | 74.2 (11.67)
  Day 7: Post-dose at 30 minutes (Period 3): number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 30 minutes (Period 3) | 67.4 (8.37) | 73.8 (11.78)
  Day 7: Post-dose at 1 hour (Period 3): number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 1 hour (Period 3) | 65.7 (7.29) | 72.9 (11.34)
  Day 7: Post-dose at 2 hours (Period 3): number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 2 hours (Period 3) | 60.9 (6.53) | 67.6 (10.22)
  Day 7: Post-dose at 4 hours (Period 3): number analyzed (Participants) | 16 | 13
  Day 7: Post-dose at 4 hours (Period 3) | 56.9 (8.19) | 67.1 (11.54)
  Baseline (Pre-dose at Day 10 (Period 4): number analyzed (Participants) | 13 | 16
  Baseline (Pre-dose at Day 10 (Period 4) | 65.5 (9.36) | 54.0 (7.77)
  Day 10: Post-dose at 15 minutes (Period 4): number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 15 minutes (Period 4) | 77.2 (11.63) | 69.3 (10.00)
  Day 10: Post-dose at 30 minutes (Period 4): number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 30 minutes (Period 4) | 77.2 (11.18) | 67.9 (9.96)
  Day 10: Post-dose at 1 hour (Period 4): number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 1 hour (Period 4) | 74.4 (10.42) | 66.4 (8.71)
  Day 10: Post-dose at 2 hours (Period 4): number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 2 hours (Period 4) | 70.2 (10.16) | 61.4 (7.71)
  Day 10: Post-dose at 4 hours (Period 4): number analyzed (Participants) | 13 | 16
  Day 10: Post-dose at 4 hours (Period 4) | 67.8 (10.21) | 58.3 (6.93)

49. Primary Outcome: Cohort 1: Area Under the Plasma Concentration-time Curve up to 30 Minutes Post- Dose (AUC[0-30])
Description: Blood samples were collected for the analysis of Pharmacokinetic (PK) parameters.
Time Frame: as for outcome 4
Population: Pharmacokinetic Population included all participants in the Full Analysis Set who had at least 1 non-missing assessment. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Hour * Picogram per Milliliter (h*pg/mL)
Arm/Group | Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) | Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference)
Number analyzed (Participants) | 29 | 29
Hour * Picogram per Milliliter (h*pg/mL) | 156.41 [135.32 to 180.79] | 162.11 [141.93 to 185.15]
Statistical Analysis 1: Comparison: Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) vs Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference); Test type: Other; Ratio of Geometric Least Squares Mean = 0.9649, 90% CI 2-sided [0.8695 to 1.0707]

50. Primary Outcome: Cohort 1: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC[0-infinity])
Description: Blood samples were collected for the analysis of Pharmacokinetic (PK) parameters.
Time Frame: At pre-dose, 3, 5, 10, 15, 20, 30, 45 minutes post-dose and at 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose on Day 1 (Period 1), Day 4 (Period 2), Day 7 (Period 3) and Day 10 (Period 4)
Population: Pharmacokinetic Population
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: h*pg/mL
Arm/Group | Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) | Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference)
Number analyzed (Participants) | 30 | 30
h*pg/mL | 5734.92 [5214.16 to 6307.68] | 4431.63 [4102.67 to 4786.97]
Statistical Analysis 1: Comparison: Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) vs Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference); Test type: Other; Ratio of Geometric Least Squares Mean = 1.2941, 90% CI 2-sided [1.1795 to 1.4199]

51. Primary Outcome: Cohort 1: Maximum Observed Plasma Concentration (Cmax)
Description: Blood samples were collected for the analysis of Pharmacokinetic (PK) parameters.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Picogram per milliliter (pg/mL)
Arm/Group | Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) | Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference)
Number analyzed (Participants) | 30 | 30
Picogram per milliliter (pg/mL) | 639.28 [578.69 to 706.20] | 518.51 [463.91 to 579.53]
Statistical Analysis 1: Comparison: Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) vs Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference); Test type: Other; Ratio of Geometric Least Squares Mean = 1.2329, 90% CI 2-sided [1.1171 to 1.3608]

52. Primary Outcome: Cohort 2: Area Under the Plasma Concentration-time Curve up to 30 Minutes Post- Dose (AUC[0-30])
Description: Blood samples were collected for the analysis of Pharmacokinetic (PK) parameters.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Hour * Picogram per Milliliter (h*pg/mL)
Arm/Group | Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) | Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference)
Number analyzed (Participants) | 30 | 29
Hour * Picogram per Milliliter (h*pg/mL) | 443.33 [374.78 to 524.43] | 467.88 [393.39 to 556.47]
Statistical Analysis 1: Comparison: Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) vs Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference); Test type: Other; Ratio of Geometric Least Squares Mean = 0.9475, 90% CI 2-sided [0.7746 to 1.1590]

53. Primary Outcome: Cohort 2: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC[0-infinity])
Description: Blood samples were collected for the analysis of Pharmacokinetic (PK) parameters.
Time Frame: as for outcome 50
Population: as for outcome 4
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: h*pg/mL
Arm/Group | Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) | Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference)
Number analyzed (Participants) | 30 | 29
h*pg/mL | 17098.45 [15794.52 to 18510.03] | 14210.59 [13339.71 to 15138.32]
Statistical Analysis 1: Comparison: Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) vs Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference); Test type: Other; Ratio of Geometric Least Squares Mean = 1.2032, 90% CI 2-sided [1.1620 to 1.2459]

54. Primary Outcome: Cohort 2: Maximum Observed Plasma Concentration (Cmax)
Description: Blood samples were collected for the analysis of Pharmacokinetic (PK) parameters.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Picogram per milliliter (pg/mL)
Arm/Group | Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) | Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference)
Number analyzed (Participants) | 30 | 29
Picogram per milliliter (pg/mL) | 1891.30 [1741.29 to 2054.24] | 1677.79 [1545.53 to 1821.37]
Statistical Analysis 1: Comparison: Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) vs Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference); Test type: Other; Ratio of Geometric Least Squares Mean = 1.1273, 90% CI 2-sided [1.0229 to 1.2423]

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 46 days [From ICF signing (Day -28) until telephonic follow-up (Day 18)]
Description: Safety Population included all participants who received at least one puff/actuation of study intervention.
Arm/Group | Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) | Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference) | Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) | Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/30 | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 12/30 | 7/30 | 16/30 | 21/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) (N=30) | Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference) (N=30) | Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) (N=30) | Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference) (N=29)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Salbutamol HFA-152a MDI 200 ug (Test) (N=30) | Cohort 1: Salbutamol HFA-134a MDI 200 ug (Reference) (N=30) | Cohort 2: Salbutamol HFA-152a MDI 800 ug (Test) (N=30) | Cohort 2: Salbutamol HFA-134a MDI 800 ug (Reference) (N=30)
Catheter site haematoma (General disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Catheter site irritation (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 9 (9) | 9 (9)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 5 (5) | 10 (10)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Hot flush (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Vessel puncture site haematoma (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/08/NCT06433908/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT06433908/SAP_001.pdf